# CLINICAL RESEARCH IN INFECTIOUS DISEASES

# STATISTICAL ANALYSIS PLAN for DMID Protocol: 23-0005

A Phase 1, Placebo-Controlled, Double-Blinded Study to Assess the Safety and Pharmacokinetics of Single Ascending Doses of EV68-228-N in Healthy Adult Volunteers

NCT06444048

Version 2.0

**DATE: 21AUG2025** 

RESTRICTED

# **STUDY TITLE**

| <b>Protocol Number Code:</b> | DMID Protocol: 23-0005 |
|---|---|
| <b>Development Phase:</b> | Phase 1 |
| Products: | EV68-228-N |
| Form/Route: | Intravenous (IV) infusion |
| Indication Studied: | Acute Flaccid Myelitis |
| Sponsor: | Division of Microbiology and Infectious Diseases |
| | National Institute of Allergy and Infectious Diseases |
| | National Institutes of Health |
| Clinical Trial Initiation Date: | 18JUN2024 |
| Clinical Trial Completion Date: | TBD |
| Date of the Analysis Plan: | 21AUG2025 |
| Version Number: | 2.0 |

This study was performed in compliance with Good Clinical Practice.

Information contained in this publication is the property of Division of Microbiology and Infectious Diseases and is confidential. This information may not be disclosed to third parties without written authorization from Division of Microbiology and Infectious Diseases. This report may not be reproduced, stored in a retrieval system or transmitted in any form or by any means - electronic, mechanical, recording or otherwise - without the prior authorization from Division of Microbiology and Infectious Diseases. This document must be returned to Division of Microbiology and Infectious Diseases upon request.

# **TABLE OF CONTENTS**

| STUDY 7 | ΓITLE | 2 |
|---|---|---|
| TABLE ( | OF CONTENTS | 3 |
| LIST OF | ABBREVIATIONS | 6 |
| 1. | PREFACE | 10 |
| 2. | INTRODUCTION | 11 |
| 2.1. | Purpose of the Analyses | 12 |
| 3. | STUDY OBJECTIVES AND ENDPOINTS | 13 |
| 3.1. | Study Objectives | 13 |
| 3.1.1. | Primary | 13 |
| 3.1.2. | Secondary | 13 |
| 3.2. | Outcome Measures | 13 |
| 3.2.1. | Primary | 13 |
| 3.2.2. | Secondary | 13 |
| 3.3. | Study Definitions and Derived Variables | 13 |
| 3.3.1. | Baseline | 13 |
| 3.3.2. | Study Day | 14 |
| 3.3.3. | Detectable Anti-Drug Antibody | 14 |
| 3.3.4. | Pharmacokinetic Parameters | 14 |
| 4. | INVESTIGATIONAL PLAN | 16 |
| 4.1. | Overall Study Design and Plan | 16 |
| 4.2. | Discussion of Study Design. | 17 |
| 4.3. | Selection of Study Population | 17 |
| 4.3.1. | Eligibility Criteria | 17 |
| 4.3.1.1. | Participant Inclusion Criteria | 17 |
| 4.3.1.2. | Participant Exclusion Criteria | 18 |
| 4.3.1.3. | Withdrawal from the Study or Discontinuation of the Study Product | 19 |
| 4.3.1.4. | Participant Replacement | 20 |
| 4.3.1.5. | Study Termination | 20 |
| 4.4. | Treatments | 20 |
| 111 | Treatments Administered | 20 |

| Table of | Contents (continued) | |
|---|---|---|
| 4.4.2. | Identity of Investigational Product(s) | 21 |
| 4.4.3. | Method of Assigning Participants to Dose Cohorts (Randomization) | 21 |
| 4.4.4. | Selection of Doses in the Study | 21 |
| 4.4.5. | Selection and Timing of Dose for Each Participant | 21 |
| 4.4.6. | Blinding | 21 |
| 4.4.7. | Prior and Concomitant Therapy | 22 |
| 4.4.8. | Treatment Compliance | 22 |
| 4.5. | Safety, Immunogenicity and Pharmacokinetic Variables | 22 |
| 4.5.1. | Safety Variables | 22 |
| 4.5.2. | Immunogenicity Variables | 23 |
| 4.5.3. | Pharmacokinetic Variables | 23 |
| 5. | SAMPLE SIZE CONSIDERATIONS | 24 |
| 6. | GENERAL STATISTICAL CONSIDERATIONS | 25 |
| 6.1. | General Principles | 25 |
| 6.2. | Timing of Analyses | 25 |
| 6.3. | Analysis Populations | 25 |
| 6.3.1. | Modified Intent-to-Treat (mITT) Population | 25 |
| 6.3.2. | Per-Protocol Population | 25 |
| 6.3.3. | Safety Population | 25 |
| 6.3.4. | Pharmacokinetics Population. | 25 |
| 6.4. | Covariates and Subgroups | 26 |
| 6.5. | Missing Data | 26 |
| 6.6. | Interim Analyses and Data Monitoring | 26 |
| 6.7. | Multicenter Studies | 26 |
| 6.8. | Multiple Comparisons/Multiplicity | 26 |
| 7. | STUDY PARTICIPANTS | 27 |
| 7.1. | Disposition of Participants. | 27 |
| 7.2. | Protocol Deviations | 27 |
| 8. | EFFICACY EVALUATION | 28 |
| 9. | SAFETY EVALUATION | 29 |
| 9.1. | Demographic and Other Baseline Characteristics | 29 |
| 911 | Prior and Concurrent Medical Conditions | 29 |

| Table of | Contents (continued) | |
|---|---|---|
| 9.1.2. | Prior and Concomitant Medications | 29 |
| 9.2. | Measurements of Treatment Compliance | 29 |
| 9.3. | Adverse Events | 29 |
| 9.3.1. | Solicited Events and Symptoms | 30 |
| 9.3.2. | Unsolicited Adverse Events | 30 |
| 9.4. | Deaths, Serious Adverse Events and other Significant Adverse Events | 31 |
| 9.5. | Pregnancies | 31 |
| 9.6. | Clinical Laboratory Evaluations | 31 |
| 9.6.1. | Clinical Laboratory Evaluations – Chemistry | 31 |
| 9.6.2. | Clinical Laboratory Evaluations - Hematology | 32 |
| 9.7. | Vital Signs and Physical Examinations | 32 |
| 9.8. | 12-Lead Standard Electrocardiogram | 33 |
| 9.9. | Prior and Concomitant Medications | 33 |
| 9.10. | Other Safety Measures | 33 |
| 10. | PHARMACOKINETICS | 34 |
| 10.1. | Summary of Pharmacokinetic Sampling and Sample Properties | 34 |
| 10.2. | Pharmacokinetic Analysis | 34 |
| 10.2.1. | Concentration Summaries | 34 |
| 10.2.2. | Pharmacokinetic Parameters | 35 |
| 11. | IMMUNOGENICITY | 36 |
| 12. | OTHER ANALYSES | 37 |
| 13. | REPORTING CONVENTIONS | 38 |
| 14. | TECHNICAL DETAILS | 39 |
| 15. | SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES | 40 |
| 16. | REFERENCES | 41 |
| 17. | LISTING OF TABLES, FIGURES, AND LISTINGS | 42 |
| APPEND | DICES | 43 |
| APPEND | DIX 1. TABLE MOCK-UPS | 44 |
| APPEND | DIX 2. FIGURE MOCK-UPS | 115 |
| APPEND | DIX 3. LISTINGS MOCK-UPS | 126 |

# **VERSION HISTORY**

| Version | Date | Change | Rationale |
|---|---|---|---|
| 1.0 | 21JUL2025 | Not Applicable | Original version |
| 2.0 | 21AUG2025 | Page 80, Table # and title updated | In v1.0, continuation of Table 34 onto next page had incorrect table number and title in error. |

# **List of Abbreviations** (continued)

# LIST OF ABBREVIATIONS

| ADA | Anti-Drug Antibodies |
|---|---|
| AE | Adverse Event |
| AFM | Acute Flaccid Myelitis |
| ALT | Alanine Aminotransferase |
| AUC | Area under the serum concentration-time curve |
| AUC <sub>0-∞</sub> | AUC from time 0 to infinity |
| AUC <sub>0-t</sub> | AUC from time 0 to time t |
| AUC <sub>0-48</sub> | AUC from time 0 to 48 hours post dose |
| AUC <sub>0-last</sub> | AUC from time 0 to the time of the last quantifiable concentration |
| BQL | Below the Quantitation Level |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| CI | Confidence Interval |
| CL | Total serum clearance |
| C <sub>max</sub> | Maximum observed serum concentration |
| CNS | Central Nervous System |
| CONSORT | Consolidated Standards of Reporting Trials |
| Cr | Creatinine |
| CRF | Case Report Form |
| CS | Clinically Significant |
| CSF | Cerebrospinal Fluid |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CV | Coefficient of Variation |
| DBP | Diastolic Blood Pressure |
| DHHS | Department of Health and Human Services |
| DMID | Division of Microbiology and Infectious Diseases, NIAID, NIH, DHHS |
| DMPA | Depot Medroxyprogesterone Acetate |

# **List of Abbreviations** (continued)

| ECG | Electrocardiogram |
|---------|----------------------------------------------|
| ECL | Electrochemiluminescence |
| ECL | Electrochemilumnescence Immunoassay |
| eCRF | Electronic Case Report Form |
| EV-D68 | Enterovirus D68 |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Amendments Act |
| GCP | Good Clinical Practice |
| GM | Geometric Mean |
| GMT | Geometric Mean Titer |
| HBV | Hepatitis B Virus |
| HCV | Hepatitis C Virus |
| Hgb | Hemoglobin |
| HIV | Human Immunodeficiency Virus |
| HLGT | High Level Group Term |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonisation |
| IgE | Immunoglobulin E |
| IV | Intravenous |
| IVIg | Intravenous Immunoglobulin |
| LARC | Long-acting Reversible Contraception |
| MAAE | Medically Attended Adverse Event |
| mAb | Monoclonal Antibody |
| MedDRA® | Medical Dictionary for Regulatory Activities |
| mITT | Modified Intent-to-Treat |
| MSD | Meso Scale Discovery |
| MRI | Magnetic Resonance Imaging |
| N | Number (typically refers to participants) |
| NCA | Noncompartmental Analysis |

# **List of Abbreviations** (continued)

| NIAID | National Institute of Allergy and Infectious Diseases, NIH, DHHS |
|---|---|
| NIH | National Institutes of Health |
| NOCMC | New Onset Chronic Medical Condition |
| NRR | "No Recorded Result" |
| PI | Principal Investigator |
| PK | Pharmacokinetics |
| Plt | Platelet |
| PSRT | Protocol Safety Review Team |
| PT | Preferred Term |
| RAMP | Rapid Antibody Manufacturing Platform |
| RNA | Ribonucleic Acid |
| SAE | Serious Adverse Event/Serious Adverse Experience |
| SAP | Statistical Analysis Plan |
| SBP | Systolic Blood Pressure |
| SD | Standard Deviation |
| SDCC | Statistical and Data Coordinating Center |
| SMC | Safety Monitoring Committee |
| SOA | Schedule of Activities |
| SOC | System Organ Class |
| t <sub>1/2</sub> | Apparent serum terminal elimination half-life |
| T bili | Total Bilirubin |
| T <sub>max</sub> | Time of the maximum observed serum concentration |
| US | United States |
| VS | Vital Signs |
| VTEU | Vaccine Treatment and Evaluation Unit |
| Vz | Volume of distribution during the terminal phase |
| WBC | White Blood Cells |
| WHO | World Health Organization |
| · | |

#### 1. PREFACE

The Statistical Analysis Plan (SAP) for "A Phase 1, Placebo-Controlled, Double-Blinded Study to Assess the Safety and Pharmacokinetics of Single Ascending Doses of EV68-228-N in Healthy Adult Volunteers" (DMID Protocol 23-0005) describes and expands upon the statistical information presented in the protocol.

This document describes all planned analyses and provides reasons and justifications for these analyses. It also includes sample tables, listings, and figures planned for the final analyses. Regarding the final analyses and Clinical Study Report (CSR), this SAP follows the International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Guidelines, as indicated in Topic E3 (Structure and Content of Clinical Study Reports), and more generally is consistent with Topic E8 (General Considerations for Clinical Trials) and Topic E9 (Statistical Principles for Clinical Trials). The structure and content of the SAP provides sufficient detail to meet the requirements identified by the FDA and ICH, while all work planned and reported for this SAP will follow internationally accepted guidelines published by the American Statistical Association and the Royal Statistical Society for statistical practice.

This document contains four sections: (1) a review of the study design, (2) general statistical considerations, (3) comprehensive statistical analysis methods for pharmacokinetics (PK) and safety outcomes, and (4) a list of proposed tables and figures. Within the table, figure, and listing mock-ups (Appendices 1, 2, and 3), references to CSR sections are included. Any deviation from this SAP will be described and justified in protocol amendments and/or in the CSR, as appropriate. The reader of this SAP is encouraged to also review the study protocol for details on conduct of the study and the operational aspects of clinical assessments.

#### 2. INTRODUCTION

Enterovirus D68 (EV-D68) is a re-emerging picornavirus associated with severe respiratory infections and neurologic diseases, such as acute flaccid myelitis (AFM). AFM is a subtype of myelitis characterized by flaccid weakness in at least one limb and magnetic resonance imaging (MRI) changes in grey matter indicating demyelination within the spinal cord. AFM occurs in ∼1% of EV-D68 infections in children with an average age of onset of 5-7 years (1, 2). A majority of AFM patients experience other symptoms of upper respiratory illness within 5-10 days prior to onset of limb weakness, and neurological sequelae typically peak within several days (≤10) of onset (1, 3). Studies have identified enterovirus antibodies in the cerebrospinal fluid of patients with AFM, and more recently EV-D68 ribonucleic acid (RNA) and protein were identified in anterior horn motor neurons of the cervical spinal cord from a 5-year-old boy who died of an AFM-like illness in 2008 (4).

AFM outbreaks have occurred worldwide and have been well characterized in the U.S., with peaks in incidence occurring in August through October every other year since 2014. The outbreak in 2014 remains the largest ever recorded EV-D68 outbreak, with 1,152 confirmed cases spanning all states except for Alaska. Over half of the hospitalized patients with respiratory disease were admitted to intensive care units, with 80% receiving supplemental oxygen, 23% requiring non-invasive ventilation, 8% requiring intubation and mechanical ventilation, and 1% died (3). Since that time, incidence has steadily increased. The biennial domestic AFM outbreaks have been associated with EV-D68 circulation, and there is now strong evidence of causality for enteroviruses and AFM. In 2020 and 2022, AFM incidence was lower than in previous years (5), likely due to social distancing measures from the ongoing COVID pandemic; however, it is likely that EV-D68 will re-emerge in years to come, leading to sustained AFM incidence.

Currently, no agent is approved in the U.S. for the treatment of severe EV-D68 infection or AFM, and the current standard of care is limited to supportive treatment and polyclonal intravenous immunoglobulin (IVIg). Commercial lots of IVIg contain varying levels of antibodies to EV-D68, and the efficacy of IVIg administration is unknown.

The human monoclonal antibody 228 was derived from patients recovering from EV-D68 infection (6). This monoclonal antibody (mAb) was found to have potent in vitro neutralizing activity against multiple clinical EV-D68 strains across multiple years (2014, 2016, and 2018 epidemic years). The 228 antibody has subsequently been produced by KBio, Inc., using genetically engineered plasmids in a Nicotiana benthamiana (tobacco plant) based rapid antibody manufacturing platform (RAMP) (product name: EV68-228-N) (7). It has been tested against EV-D68 in vitro and in vivo and has demonstrated therapeutic effects when administered soon after the onset of neurological symptoms in a murine model of EV-D68 infection.

In a murine neurologic model of infection that mimics human AFM, mAb EV68-228-N treatment eliminated detectable virus from the blood within 24 hours of administration; improved survival and neurologic disease when given up to 48 hours after infection; and improved clinical response when given as late as 72 hours after infection. In a separate in vivo murine model of EV-D68 induced AFM, mAb EV68-228-N treatment effectively prevented progression of paralysis and improved histopathologic evidence of disease in tissues of the central nervous system (CNS) when treatment was initiated after the onset of limb weakness; most critically, EV68-228-N treatment conferred a protective effect on CNS motor neurons following EV-D68-infection induced paralysis. These data support the hypothesis that mAb EV68-228-N is a potent neutralizing antibody in vivo and can result in clinical improvement in murine models of EV-D68 infection, even when administered after the onset of neurologic disease (7).

While the pathogenesis of AFM is incompletely understood, targeting the replicating virus with a neutralizing monoclonal antibody appears to be a reasonable next step based on recent human data. Vogt, Wright, and Hickey reported on a 5-year-old boy who died of an AFM-like illness in 2008 (4). EV-D68 was detected in the cerebrospinal fluid (CSF) and using preserved formalin-fixed and paraffin-embedded autopsy tissue, the authors were able to detect EV-D68 RNA and protein in anterior horn motor neurons and their axons using in situ hybridization and immuno-histochemistry. In addition, Vogt et al identified CD8+ T-cell and CD68+ macrophage infiltration in EV-D68-infected regions along with up-regulated inflammatory gene transcripts in inflamed tissues. Not only do these data support the causal association between EV-D68 and AFM, but they also support the hypothesis that the clinical presentation of AFM includes a combination of the direct effects of viral infection of spinal cord motor neurons and damage resulting from local inflammation. Taken together, the data supports ongoing efforts to develop antiviral and neutralizing monoclonal antibody treatment options that may aid in viral clearance and possible immunomodulation.

Given the therapeutic potential of EV68-228-N and the exceptional safety profile of fully human monoclonal antibodies, further development is warranted. This Phase 1 clinical trial will evaluate the safety and PK of EV68-228-N in healthy adult volunteers to support future evaluations of its efficacy as a treatment for AFM in pediatric patients.

# 2.1. Purpose of the Analyses

These analyses will assess the safety and PK of EV68-228-N after a single IV infusion in healthy adult male and female volunteers. Safety and PK data from the Phase 1 study of EV68-228-N will be used to support identification of a target dose for future efficacy trials in AFM patients.

#### 3. STUDY OBJECTIVES AND ENDPOINTS

# 3.1. Study Objectives

#### **3.1.1. Primary**

• To evaluate the safety of a single IV infusion of either 3, 10, or 30 mg/kg of EV68-228-N when administered to healthy adults.

#### 3.1.2. Secondary

- To characterize the PK of single ascending doses of EV68-228-N for approximately four months following the infusion.
- To measure the occurrence of Anti-Drug Antibodies (ADAs) elicited following a single IV infusion of EV68-228-N in healthy adults.

#### 3.2. Outcome Measures

#### **3.2.1. Primary**

- Proportion of participants experiencing solicited adverse events (AEs) through 48 hours post-infusion.
- Proportion of participants experiencing unsolicited AEs including clinical and laboratory AEs through Day 29.
- Proportion of participants experiencing serious AEs (SAEs), medically attended AEs (MAAEs), and new onset chronic medical conditions (NOCMCs) through the end of the study.

#### 3.2.2. Secondary

After a single IV infusion of EV68-228-N:

- EV68-228-N concentrations in serum will be determined with a validated assay. The PK parameters will be estimated based on the concentration-time data, including area under the serum concentration-time curve (AUC) from time 0 to infinity (AUC₀-∞), AUC from time 0 to 48 hours post dose (AUC₀-48), AUC from time 0 to the time of the last quantifiable concentration (AUC₀-last), maximum observed serum concentration (C<sub>max</sub>), time of the C<sub>max</sub> (T<sub>max</sub>), apparent serum terminal elimination half-life (t₁/2), total serum clearance (CL), and volume of distribution during the terminal phase (Vz) calculated from serum EV68-228-N levels.
- Incidence of anti-EV68-228-N antibodies as measured by the proportion of participants with detectable anti-EV68-228-N antibodies in serum.

# 3.3. Study Definitions and Derived Variables

#### 3.3.1. Baseline

For clinical laboratory and serological and electrocardiogram (ECG) measurements, the last value recorded prior to administration of study drug will be considered as baseline. For vital signs (VS) measurements, generally the last value recorded prior to administration of study drug will also be considered as baseline, but

if repeat measurements are collected at the baseline visit, the rules in Section 9.7 will be used to determine which result will be used as the actual baseline value.

Baseline height was obtained at screening. Weight was obtained at both screening and Day 1 prior to dosing; the baseline weight will be the one obtained at Day 1. Baseline body mass index (BMI) will be calculated using the height measure at screening and the weight measure at Day 1. Age will be based on age at the time of enrollment.

#### **3.3.2. Study Day**

Study day will primarily be used in listings to refer to the timing of assessments and events relative to study drug administration. The day that the administration of study drug is received is considered Study Day 1 for all participants. The day prior to the administration of study drug is considered Study Day -1; there is no Study Day 0.

Participation for an individual participant will be approximately four to six months, which includes a 1 to 28-day screening period, infusion on Day 1, and follow-up visits on Day 2, 3, 8, 15, 29, 61, 91, and 121.

## 3.3.3. Detectable Anti-Drug Antibody

There are three steps in the Meso Scale Discovery (MSD) Electrochemiluminescent (ECL) assay: screening assay, confirmatory assay, and titer assay. The screening assay will have qualitative results of negative (NEG), potential positive screening (PPS) and no recorded result (NRR).

An ADA confirmatory assay will be performed for specimens with PPS screening results. The result of the confirmatory assay is qualitative, NEG, NRR, or positive (POS).

A detectable ADA is defined when the confirmatory assay result is POS.

#### 3.3.4. Pharmacokinetic Parameters

AUC<sub>0- $\infty$ </sub> is defined as the AUC from the time of dosing extrapolated to time infinity based on the last observed concentration (C<sub>last</sub>) and the elimination rate constant ( $\lambda z$ ), where C<sub>last</sub> is defined as the last observed positive concentration above the lower limit of quantitation (LLOQ) and  $\lambda z$  is defined as the first-order rate constant associated with the terminal (log-linear) portion of the curve describing the rate of elimination from serum. Estimated by linear regression of time vs. log concentration. AUC<sub>0- $\infty$ </sub> will be computed by adding AUC<sub>0-last</sub> to an area extrapolated by C<sub>last</sub> divided by  $\lambda z$ , as shown below:

$$AUC_{0-\infty} = AUC_{0-last} + \frac{C_{last}}{\lambda_z}$$

AUC<sub>0-last</sub> is defined as the AUC from the time of dosing to the time of the last quantifiable concentration above the LLOQ based on observed concentrations.

AUC<sub>0-48</sub> is defined as the AUC from the time of dosing to the time of the last quantifiable concentration above the LLOQ up to and including the nominal 48 hr time point based on observed concentrations.

Maximum serum concentration ( $C_{max}$ ) is defined as the maximum observed concentration, occurring the time of maximal serum concentration ( $T_{max}$ ), in serum following the first dose of EV68-228-N.

T<sub>max</sub> is defined as the time at which the maximum observed serum concentration occurs. Because non-steady-state data is collected, the entire curve is considered. If the maximum observed concentration is not unique, then the first maximum is used.

The terminal elimination half-life ( $t_{1/2}$ ) is defined as the time it takes serum concentrations to reduce by 50% during the terminal elimination phase and will be estimated by the natural logarithm of 2 (ln(2)) divided by  $\lambda z$ .

Total serum clearance (CL) is defined as the total clearance and represents a volume that is cleared of the molecule of interest per hour. It will be calculated as the dose divided by the  $AUC_{0-\infty}$ , as shown below:

$$CL = \frac{Dose}{AUC_{0-\infty}}$$

The volume of distribution during the terminal phase  $(V_z)$  is defined as the theoretical volume that the total amount of the molecule of interest would occupy if uniformly distributed at the concentration observed in serum. If the terminal phase has been adequately captured, this value should approximate the volume of distribution at steady state and is calculated as shown below:

$$V_z = \frac{Dose}{\lambda_z \times AUC_{0-\infty}} = \frac{CL}{\lambda_z}$$

#### 4. INVESTIGATIONAL PLAN

# 4.1. Overall Study Design and Plan

This is a Phase 1, randomized, placebo-controlled, double-blinded study to assess the safety and PK of single IV administrations of EV68-228-N in healthy adult volunteers.

Three doses (3, 10 and 30 mg/kg) of EV68-228-N will be evaluated in three separate, sequential cohorts (N = 12, each cohort) in this single dose escalation study. The cohorts will be randomized in a 5:1 randomization scheme for EV68-228-N and placebo. The first two participants in each cohort will serve as sentinels. Sentinel participants may be located at different sites. Sentinel safety data will be collected through Day 3 before submitting to the Protocol Review Safety Team (PSRT) for review. The PSRT is comprised of the Principal Investigator (PI), the DMID Medical Monitor, and the DMID Medical Officer.

Data to be reviewed will include clinical data collected from Visits 1, 2 and 3, the results of laboratory testing conducted at these visits, solicited AEs and the passive reporting of AEs through Day 3. From the time of infusion of the sentinels to at least 48 hours after infusion, no new participants will be given study product or placebo, but screening may continue. If no safety signal is detected in the sentinel group, and after approval from the DMID Medical Monitor, the remaining 10 participants in the cohort will be dosed following the overall 5:1 randomization scheme.

All participants will be actively monitored for AEs and safety laboratory data following dosing through Day 8. Data will be reviewed by the PSRT and discussed with the SMC for their concurrence before advancing to the next cohort. Electronic review of the safety data by the SMC is required prior to the cohort dose escalation when halting rules are met or there are any safety concerns.

Assuming no safety concerns are identified after review of the first cohort safety data through Day 8, enrollment of Cohort 2 will begin. The dose of EV68-228-N will be increased to 10 mg/kg for the second cohort. The same sentinel design and safety plan will be used to evaluate sentinel participants in Cohort 2 and determine whether to enroll the remaining participants in Cohort 2. In addition, the same sentinel design and safety plan will be used for Cohort 3, which will evaluate the 30 mg/kg dose.

Following informed consent, participants will be screened for eligibility, including medical history, physical examination, weight and height measurements, VS, screening laboratory tests, and a 12-lead ECG. Within 28 days of screening, eligible participants will be seen at the clinical research unit (Day 1) and be randomized to receive either a single IV dose of EV68-228-N or placebo (formulation buffer alone). Participants will remain in the unit for at least 5 hours following infusion and return for assessments on Day 2 and Day 3. Participants will have subsequent follow-up clinic visits on Days 8, 15, 29, 61, 91, and 121.

Participants will be monitored and assessed for safety and the incidence of AEs at all visits beginning with the dosing visit. An electronic memory aid will be utilized from Day 1 through Day 3 to assist with collecting solicited AEs. Safety laboratory studies will be collected at screening and on Days 1, 2, 3, 8, and 29. Concomitant medications taken 28 days before and after dosing will be recorded.

PK samples will be collected prior to infusion, at the end of infusion, at 1, 3, 5, 24 and 48 hours after end of infusion; and on Days 8, 15, 29, 61, 91, and 121. The single dose PK parameters to be estimated include  $C_{max}$ ,  $T_{max}$ , -  $AUC_{0-48}$ ,  $AUC_{0-last}$ , and  $AUC_{0-\infty}$ ,  $t_{1/2}$ , CL, and Vz. PK parameters will be calculated from serum EV68-228-N levels measured using a validated ECL assay performed by PPD, Inc..

Samples for serum levels of anti-EV68-228-N antibodies will be collected prior to infusion on Day 1 and on Days 8, 15, 29, 61, 91 and 121.

A sample will be collected pre-infusion on Day 1 for hypersensitivity testing in the event that the participant experiences an infusion reaction. These baseline samples will only be analyzed in the event of a hypersensitivity reaction related to the infusion. If a participant experiences anaphylaxis or an anaphylactoid event related to the infusion, three additional samples will be collected: 1) during onset, 2) 2 or more hours after onset, and 3) after resolution of symptoms.

The study dosing plan is shown in Table 1.

# 4.2. Discussion of Study Design

This is a Phase 1, randomized, placebo-controlled, double-blinded study to assess the safety and PK of a single IV infusion of EV68-228-N in healthy adult volunteers. All participants will be actively monitored for solicited AE following infusion through Day 3 and clinical and safety laboratory data following dosing through Day 8. Three doses (3, 10 and 30 mg/kg) of EV68-228-N will be evaluated in three separate, sequential cohorts in this single dose escalation study. The cohorts will be randomized in a 5:1 randomization scheme. All placebo participants are analyzed jointly across cohorts. The first two participants in each cohort will serve as sentinels. Sentinel participants may be located at different sites.

# 4.3. Selection of Study Population

As this is the first time EV68-228-N will be tested in humans, the study population will be comprised of healthy males and non-pregnant, non-lactating females, ages 18-49 years inclusive at the time of consent, regardless of religion, sex, or ethnic background, who meet all of the inclusion and none of the exclusion criteria. The eligibility criteria apply only to enrollment of participants into the study. The focus population should reflect the community at large at the site. Participant Inclusion and Exclusion Criteria must be confirmed by a study clinician licensed to make medical diagnoses. No exemptions are granted on Subject Inclusion/Exclusion Criteria in DMID-sponsored studies. Questions about eligibility will be directed toward the DMID Medical Officer.

## 4.3.1. Eligibility Criteria

#### 4.3.1.1. Participant Inclusion Criteria

- 1. Provides written informed consent prior to initiation of any study procedures.
- 2. Is able to understand and agrees to adhere to planned study procedures and is available for all study visits.
- 3. Adult volunteers 18 to 49 years of age, inclusive.
- 4. Females who are of childbearing potential must agree not to become pregnant.

<sup>1</sup> Not of childbearing potential includes post-menopausal females (defined as no menses for at least 12 months without an alternative medical cause for amenorrhea) or surgically sterile females with documented history of hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure® placement.

- 5. Females who have sexual intercourse with male partners must agree to use at least one acceptable form of contraception for the duration of the study<sup>2,3</sup>.
  - <sup>2</sup> Acceptable methods of birth control include long-acting reversible contraception (LARC), combined pill, progestin-only pill, hormone-releasing transdermal patch or vaginal ring, and depot medroxyprogesterone acetate (DMPA) injection. Participants who choose to use a licensed hormonal product should use them for a minimum of 28 days prior to study infusion. True sexual abstinence or a monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the participant's first infusion are also acceptable contraceptive methods.
  - <sup>3</sup> Participants who report practicing true abstinence, defined as no heterosexual vaginal-penile intercourse, need to practice true abstinence at all times during the study. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and the withdrawal method are not acceptable methods of contraception.
- 6. Females of childbearing potential must agree to not donate ova or oocytes during the study.
- 7. Participant is in good health<sup>4</sup>.
  - <sup>4</sup> Good health is defined by the absence of a medical condition described in the exclusion criteria. If the participant has another current, ongoing medical condition, the condition cannot meet any of the following criteria: (1) was first diagnosed within 3 months of enrollment with a clinically significant condition, in the opinion of investigator that has worsened within 3 months of enrollment; (2) had non-elective surgery, clinically significant medical procedure, or hospitalization within 3 months of enrollment; (3) received new prescription for systemic medication within 30 days of enrollment, unless the new prescription is in the same class of agent or a transition from generic to/from brand name equivalent; or (4) takes medication that may pose a risk to participant's safety or impede assessment of adverse events or study endpoints if they participate in the study.
- 8. Must agree to refrain from donating blood or blood products<sup>5</sup> during the study.
  - <sup>5</sup> This includes whole blood cells, red blood cells, platelets, plasma, and plasma derivatives collected and donated outside of the study blood draws.
- 9. Body mass index (BMI) 18 kg/m<sup>2</sup> to 32 kg/m<sup>2</sup>, inclusive, and a weight of 125 kg or less at time of screening.
- 10. Must have adequate venous access for intravenous (IV) infusion and blood sampling.

#### 4.3.1.2. Participant Exclusion Criteria

All participants meeting any of the exclusion criteria at baseline will be excluded from study participation.

- 1. Positive pregnancy test at screening or prior to infusion.
- 2. Female participant who is lactating.
- 3. Presence of significant psychiatric condition, that in the opinion of the site PI or appropriate sub-investigator, precludes study participation.
- 4. History of drug abuse or alcohol abuse within 6 months of enrollment that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation.
- 5. Has a significant acute illness (with or without fever), as determined by the site PI or appropriate sub-investigator, within 72 hours prior to infusion<sup>1</sup>.
  - <sup>1</sup>If the participant meets all other eligibility criteria, they may be enrolled and dosed once they meet this eligibility criterion. If the illness resolves within the 28-day screening window, they do not need to be rescreened, otherwise they will need to be rescreened.
- 6. Currently enrolled in or plans to participate in another clinical trial with an investigational agent that will be received during the study-reporting period.
- 7. Has a history of significant hypersensitivity, intolerance, or allergy to any drug compound, vaccine, food, or other substance, unless approved by the Investigator (or designee)<sup>2</sup>.

- 8. Any history of an infusion reaction to any biologic product.
- 9. Receipt of a monoclonal antibody in the 180 days prior to infusion.
- 10. Receipt of a blood product within 120 days prior to infusion.
- 11. Received any live-attenuated vaccine in the 28 days prior or any other vaccine in the 14 days prior to infusion.
- 12. Has used any prohibited medication within 30 days prior to Day 1 or plans to use prohibited medication<sup>3</sup> during the study.

<sup>3</sup>Prohibited medications include systemic immunosuppressive drugs, immune modulators (except acetaminophen or non-steroidal anti-inflammatory drugs), oral corticosteroids, and systemic anti-neoplastic agents. Topical, inhaled, and intranasal steroids, as well as topical anti-neoplastic agents are acceptable.

13. Has clinically significant findings<sup>4</sup> on 12-lead electrocardiogram.

<sup>4</sup>Clinical significance will be determined by a cardiologist. Examples of findings that will lead to exclusion are significant left ventricular hypertrophy, right or left bundle branch block, advanced A-V heart block, non-sinus rhythm (excluding isolated premature atrial contractions), pathologic Q wave abnormalities, significant ST-T wave changes, and prolonged QTc interval. Long QT interval is defined in males as a median QTcB greater than 450 msec or in females as a median QTcB greater than 460 msec (Bazett's correction) at screening.

14. Abnormal vital signs (Grade 1 or higher)<sup>5</sup> at screening or on Day 1.

<sup>5</sup> Grade 1 or higher is equivalent to:

Systolic blood pressure (SBP) > 140 mmHg or < 85 mmHg Diastolic blood pressure (DBP) > 90 mmHg Oral temperature  $\geq$  38.0°C (100.4°F)

15. Abnormal laboratory results<sup>6</sup> that are Grade 1 or worse at screening based on the Toxicity Tables.

<sup>6</sup>Creatinine, alanine transaminase (ALT), hemoglobin (Hgb), platelets (PLT), white blood cell count (WBC), and total bilirubin (T bili).

<sup>7</sup>Laboratory studies can be repeated once if an alternative, transient etiology for abnormal laboratory values is identified.

- 16. Known, current human immunodeficiency virus (HIV), hepatitis B Virus (HBV), or hepatitis C virus (HCV) infection.
- 17. Has any medical disease or condition<sup>8</sup> that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation<sup>9</sup>.

<sup>8</sup>Medical conditions include, but are not limited to, kidney disease with creatinine clearance < 90 mL/min/1.73 cm² (CKD-EPI method); known active liver disease including steatosis; ischemic heart disease, clinically significant cardiac conduction disorder, arrythmia requiring treatment, congenital long QT syndrome, uncompensated heart failure; diabetes requiring insulin; neuropathy or myopathy; and malignancy (not including squamous cell skin cancer, basal cell skin cancer, or cervical low-grade squamous intraepithelial lesions).

<sup>9</sup>Participation may be precluded due to safety concerns or inability to adequately evaluate clinical trial endpoints.

#### 4.3.1.3. Withdrawal from the Study or Discontinuation of the Study Product

Participants may voluntarily withdraw their consent for study participation at any time without penalty or loss of benefits to which they are otherwise entitled.

An investigator may also withdraw a participant prior to receiving the study product or after receiving the study product for any reason. Follow-up safety evaluations will be conducted, if the participant agrees. If a

<sup>&</sup>lt;sup>2</sup>Sensitivity to glycine, citric acid, trisodium citrate, sorbitol, or polysorbate 80 (components of the study product) is exclusionary.

participant withdraws or is withdrawn prior to completion of the study, the reason for this decision must be recorded in the case report forms (CRFs).

The reasons might include, but are not limited to the following:

- Participant becomes pregnant prior to infusion.
- Participant no longer meets eligibility criteria (e.g., develops acute febrile illness on Day 1 prior to infusion).
- Participant meets individual halting criteria.
- Participant becomes non-adherent.
- Participant develops a medical disease or condition, or new clinical finding(s) for which continued
  participation, in the opinion of the investigator might compromise the safety of the participant,
  interfere with the participant's successful completion of this study, or interfere with the evaluation of
  responses.
- Participant is lost to follow-up.
- Determined by a physician's discretion to require additional therapy not indicated in the protocol to ensure participant's health and well-being.

If the participant consents, every attempt will be made to follow all AEs and pregnancies through resolution. The investigator should be explicit regarding study follow-up (e.g., safety follow-up) that might be carried out. The procedures that collect safety data for the purposes of research must be inclusive in the original informed consent or the investigator may seek subsequent informed consent using an IRB/IEC-approved consent form with the revised procedures.

The investigator will inform the participant that already collected data will be retained and analyzed even if the participant withdraws from this study.

#### 4.3.1.4. Participant Replacement

Participants who withdraw, or are withdrawn from this study, or are lost to follow-up after signing the informed consent form (ICF) and receiving an infusion will not be replaced. Participants who withdraw, or are withdrawn from this study, or are lost to follow-up after signing the ICF but before infusion may be replaced.

#### 4.3.1.5. Study Termination

If the study is prematurely terminated by the sponsor, any regulatory authority, or the investigator for any reason, the investigator will promptly inform the study participants and assure appropriate therapy or follow-up for the participants, as necessary. The investigator will provide a detailed written explanation of the termination to the IRB.

## 4.4. Treatments

#### 4.4.1. Treatments Administered

Participants will receive a single IV dose of either study product or placebo. Infusions will be administered over approximately 15 minutes or 30 minutes, depending upon the volume of the infusion, in the absence of infusion reactions or non-drug, infusion related safety issues; longer infusion times will be permitted. All infusions must be completed within 4 hours of compounding.

## 4.4.2. Identity of Investigational Product(s)

The EV68-228-N mAb is produced by expression of genetically engineered plasmids in a *Nicotiana* benthamiana based RAMP using proprietary plasmid vectors with plant viral sequences to reduce cost and improve the speed of production. The use of an engineered strain of N. benthamiana in which the plant specific glycosyltransferases,  $\alpha 1,3$  fucosyltransferase and  $\beta 1,2$  xylosyltransferase, are mutated allows the RAMP-produced mAbs to have highly homogenous mammalian N-glycans and mitigates the potential for immunogenicity caused by carryover of plant glycans. See the IB for additional information regarding product manufacturing (7).

KBio uses an internal nomenclature system for identification of investigational products; the internal KBio nomenclature for EV68-228-N is "KB13A.1.1". This identification number will appear on the Certificate of Analysis as well as product labeling.

#### 4.4.3. Method of Assigning Participants to Dose Cohorts (Randomization)

Enrollment/randomization will be performed through the enrollment module in the electronic data capture system, maintained by the Statistical and Data Coordinating Center (SDCC). Eligible participants in three dose escalating cohorts will be randomized in a 5:1 ratio to receive either EV68-228-N or placebo. The randomization is based on a variable blocked scheme to provide an approximately balanced allocation to the Dose Cohorts during the study.

### 4.4.4. Selection of Doses in the Study

Single ascending doses (3, 10, and 30 mg/kg) of EV68-228-N had been selected for this study based on the favorable safety and tolerability profile observed in the nonclinical studies (7, 8, 9, 10, 11, 12).

#### 4.4.5. Selection and Timing of Dose for Each Participant

This trial will evaluate the PK and safety of single ascending doses (3, 10, and 30 mg/kg) of EV68-228-N administered as IV infusion on Day 1. Dosing for each cohort will begin with two sentinel participants. There will be a minimum of 2 days of observation following dosing of the sentinels before dosing of additional participants in each cohort is authorized.

## 4.4.6. Blinding

All investigative site personnel, study volunteers, DMID personnel will remain blinded through database lock, with the exception of an unblinded pharmacist/verifier at the research site, an unblinded SDCC biostatistician, and a DMID manager responsible for PK sample storage. The randomization scheme will be provided to the unblinded research pharmacist at the site, who will perform dose preparation, and a pharmacy verifier who will not participate in dose preparation. The pharmacy personnel at the site will not be involved in study-related assessments or have participant contact for data collection following study drug administration. The study staff participating in the administration of study product and assessment of the participants will not be aware of the administered contents of the IV infusion in the randomized arms of the study. Study drugs will be diluted in normal saline, and they will look identical to placebo in the IV infusion bag so the study staff and the participant will not be able to determine whether placebo or active drug are being administered. The label on the IV infusion bag will not have information that can identify the contents. Individual samples are barcoded, and the barcode includes information that can match the sample to the volunteer identification number, aliquot number, treatment cohort and collection time point. The SMC will receive blinded data in aggregate and presented by cohort. The SMC may review unblinded data prepared by an unblinded biostatistician in the closed session only.

## 4.4.7. Prior and Concomitant Therapy

Medications taken before or after dosing will be reported as Prior Medications or Concomitant Medications, respectively.

Administration of any medications, therapies, or vaccines will be recorded on the appropriate data collection form. Concomitant medications recorded will include all current medications and medications taken within 28 days prior to signing the informed consent and during the study period. Medications reported in the electronic case report form (eCRF) are limited to those taken within 28 days prior to the study drug administration or taken through the study. Prescription and over-the-counter drugs will be included as well as herbals, vitamins, and supplements.

Systemic medications that might interfere with the evaluation of the investigational product should not be used unless absolutely necessary. A participant will be withdrawn for use of excluded medications. Medications in this category include the prohibited medications per the Participant Exclusion Criteria (Section 4.3.1.2). Prohibited medications include systemic immunosuppressive drugs, immune modulators (except acetaminophen or non-steroidal anti-inflammatory drugs), oral corticosteroids, and systemic anti-neoplastic agents. Topical, inhaled, and intranasal steroids, as well as topical anti-neoplastic agents are acceptable.

## 4.4.8. Treatment Compliance

All participants were to receive a single dose of study product administered in the clinic.

# 4.5. Safety, Immunogenicity and Pharmacokinetic Variables

The following section describes the safety and PK endpoints of the study. As this study is a Phase 1 clinical trial in healthy adult participants, there will be no assessment of drug efficacy. For a detailed SOA, refer to Table 2. Refer to Section 3 for a list of primary, secondary objectives and endpoints.

#### 4.5.1. Safety Variables

Safety will be assessed through the evaluation of AEs, SAEs, vital signs, ECGs, and clinical safety laboratory data as outlined in the SOA.

Solicited AEs will be summarized by severity for each day post administration (Days 1 - 3) and as the maximum severity over all 3 days. If the AE is still ongoing after Day 3, the time point will be defined as "Ongoing after Day 3". Additionally, solicited AEs will be analyzed using standard techniques, such as exact confidence intervals (CIs), to summarize the proportion of participants reporting each symptom.

Unsolicited AEs will be collected from the time of infusion through Day 29.

Unsolicited AEs will be coded by MedDRA for Preferred Term (PT), High Level Group Term (HLGT) and System Organ Class (SOC). SAEs, MAAEs and NOCMCs will be collected from the time of infusion through end of study. The numbers of SAEs, MAAEs, and NOCMCs will be reported by detailed listings showing the event description, MedDRA PT, HLGT and SOC, relevant dates (product administration and AEs), severity, relatedness, and outcome for each event. Non-serious unsolicited AEs will be summarized as number and percentage of participants reporting at least one event in each MedDRA PT, HLGT and SOC, cross tabulated by severity and relationship to study product. Additionally, the proportion of participants and exact 95% CIs of AEs in aggregate and by MedDRA categories will be computed.

Clinical laboratory and hematology measurements will be collected at Screening, pre-infusion on Day 1, and Days 2, 3, 8, and 29. ECG measurements will be collected at Screening, pre-infusion and 1-hour post-infusion

on Day 1, and Day 2. VS measurements will be collected at Screening, pre-infusion, post-infusion, and 1-hour post-infusion on Day 1, and Days 2, 3, 8, 15, and 29. Clinical laboratory, ECG, and VS results will be assessed at baseline and each post-dose time point collected, using the toxicity grading scales in Table 5. For continuous parameters, change from baseline will also be summarized for all post-dose time points. For definitions of baseline, refer to Section 3.3.1.

#### 4.5.2. Immunogenicity Variables

In this study, the immunogenicity data are measuring the anti-drug response. A validated ECL assay will be performed on samples collected approximately within 15 minutes prior to the infusion on Day 1 and at Days 8, 15, 29, 61, 91 and 121 (with corresponding windows) for serum levels of anti-EV68-228-N antibodies. To measure ADA, anti-drug antibodies will be captured by EV68-228-N and detected with labeled EV68-228-N (e.g., biotin) followed by standard detection (e.g., streptavidin -SULFO-TAG).

#### 4.5.3. Pharmacokinetic Variables

Serum EV68-228-N concentrations: The MSD ECL assay will be performed on samples collected approximately 15 minutes prior to infusion; at end of infusion ( $\pm$ 5 minute window); 1-, 3-, and 5-hours after end of infusion, within a  $\pm$ 15 minute window; 24 and 48-hours after the end of the infusion (within a  $\pm$ 3-hour window) and on Days 8, 15, 29, 61, 91, and 121 (within  $\pm$ 1-, 2-, 3-, 7-, 14-, and 14-day window, respectively). An EV68-228-N anti-idiotype antibody will be used in the assay to capture EV68-228-N and this will be detected with an anti-Human IgG (Fc)-biotin antibody, secondary detection is Streptavidin SULFO-TAG.

PK parameters will be estimated based on the time-concentration data through a non-compartmental analysis. Estimated total serum PK parameters will include the following:

- AUC<sub>0-∞</sub>: Area under the concentration time-curve from time 0 extrapolated to infinity
- AUC<sub>0-last</sub>: Area under the concentration time-curve from time 0 to the last concentration above the lower limit of quantitation
- AUC<sub>0-48</sub>: Area under the concentration time-curve from time 0 to 48hrs
- C<sub>max</sub>: Maximum concentration
- T<sub>max</sub>: Time of maximum concentration
- $t_{1/2}$ : Apparent terminal elimination half-life
- CL: Total serum clearance
- V<sub>z</sub>: Volume of Distribution during terminal phase

Refer to Section 3.3.4 for parameter definition.

#### 5. SAMPLE SIZE CONSIDERATIONS

As a Phase 1, first-in-human study, the number of participants was chosen principally on feasibility and using a 5:1 randomization scheme. Thus, three cohorts of 10 participants each (n=30) and 6 placebo recipients (total N=36) are proposed. With 10 participants in each cohort receiving study product, the chance of observing at least one AE of probability 20% or more is approximately 89.3% (see Table 3). Therefore, if no AEs of a given type occur in an active dose group, we can be relatively confident that they will occur in fewer than 20% of people once the treatment is implemented.

PK parameters are not a primary outcome of the study, so it has not been powered for this, however with a sample size of 10 participants per dose level, assuming the pharmacokinetics are not dose proportional, a parameter with a coefficient of variation of 120% or less has a 90% chance to be observed within 80% and 120% of the geometric mean.

#### 6. GENERAL STATISTICAL CONSIDERATIONS

# **6.1.** General Principles

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, SD, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures.

In general, all data will be listed, sorted by treatment, cohort, and participant, and when appropriate by visit number within participant. All summary tables will be structured with a column for each treatment in the order (3, 10, 30 mg/kg EV68-228-N, and Placebo) and will be annotated with the total population size relevant to that table/treatment, including any missing observations. In some safety tables, all participants who received active product (3, 10, 30 mg/kg EV68-228-N) will also be summarized together.

# **6.2.** Timing of Analyses

The final analysis will be performed after the final data lock, and CSR completed when all primary safety endpoint data and all secondary immunogenicity and pharmacokinetics endpoint data are available and received by the SDCC.

# 6.3. Analysis Populations

#### **6.3.1.** Modified Intent-to-Treat (mITT) Population

The mITT population includes all participants who received at least a partial dose of study product and contributed both pre- and at least one post-dose venous blood sample for immunogenicity testing for which valid results were reported. Descriptive summaries of immunogenicity data will be presented for the mITT population.

#### **6.3.2.** Per-Protocol Population

In the final analysis, protocol deviations will be reviewed to determine which protocol deviations may affect the analysis.

The per protocol population includes all participants in the mITT subset with the following exclusions:

- Data from all available visits for participants found to be ineligible at baseline.
- Data from all visits subsequent to the protocol deviations that are considered to affect the science.
- Data from any visit that occurs substantially out of window.

#### 6.3.3. Safety Population

Safety Population is defined as any participant who received all or part of the study product. Summaries and analysis of safety data will be presented for the safety population.

#### 6.3.4. Pharmacokinetics Population

The PK population will consist of participants in the Safety Population who have at least one evaluable serum PK sample for the estimation of  $C_{max}$  or  $AUC_{0-\infty}$  and received a full dose. This set will be used to assess the

PK endpoints. Any participants or data values excluded from this analysis set will be identified, along with their reason for exclusion. Participants receiving placebo are excluded from PK analysis.

# 6.4. Covariates and Subgroups

The protocol does not define any formal subgroup analyses, and the study is not adequately powered to perform subgroup analyses.

# 6.5. Missing Data

All attempts will be made to collect all data per protocol. As missing data are expected to be minimal, no imputation will be performed for missing values. Any data point that appears to be erroneous or inexplicable based on clinical judgment will be investigated as a possible outlier.

# 6.6. Interim Analyses and Data Monitoring

Not applicable.

## **6.7.** Multicenter Studies

Data will be pooled across all clinical sites. Center effects are not anticipated because the sites are using standardized procedures for infusion and assessment of solicited and unsolicited AEs, and the assessment of immunogenicity and PK endpoints will be performed at central laboratories.

# **6.8.** Multiple Comparisons/Multiplicity

This is a Phase 1 study with multiple primary endpoints. Because analyses of primary endpoints are descriptive rather than hypothesis tests, no adjustments for multiple testing are planned.

#### 7. STUDY PARTICIPANTS

# 7.1. Disposition of Participants

Table 9 will present a summary of the reasons that participants were screened but not enrolled.

The composition of analysis populations, including reasons for participant exclusion, by Dose Cohort is presented in Table 7. Individual participants who were excluded from analysis populations are presented in Listing 5.

The disposition of participants in the study will be tabulated by Dose Cohort (Table 6). The table shows the total number of participants screened, enrolled, receiving treatment, completed final blood draws, terminated from study follow-up and the number completing the study.

A flowchart showing the disposition of study participants will be included (Figure 1). This figure will present the number of participants screened, enrolled, lost to follow-up, and analyzed, by treatment arm.

A listing of participants who terminated from study follow-up and the reason will be included in Listing 2.

#### 7.2. Protocol Deviations

A summary of participant-specific protocol deviations will be presented by the reason for the deviation, the deviation category, and Dose Cohort for all participants (Table 4). Deviations that are considered major deviations will be reviewed for possible exclusion from the Per-Protocol Population. All participant-specific protocol deviations and non-participant specific protocol deviations will be included in Appendix 3 as data listings (Listing 3 and Listing 4, respectively).

# 8. EFFICACY EVALUATION

Not applicable.

#### 9. SAFETY EVALUATION

# 9.1. Demographic and Other Baseline Characteristics

Summaries of age, sex, ethnicity, and race will be presented by Dose Cohort overall and by site (Table 10, Table 11, Table 12, and Table 13). Ethnicity is categorized as Hispanic or Latino, or not Hispanic and not Latino. In accordance with NIH reporting policy, participants may self-designate as belonging to more than one race or may refuse to identify a race, the latter reflected in the CRF as "No" to each racial option.

Individual participant listings (Appendix 3) will be presented for all demographics (Listing 6).

#### 9.1.1. Prior and Concurrent Medical Conditions

All current illnesses and past pre-existing medical conditions will be MedDRA® coded using MedDRA dictionary version 27.1 or higher version.

Summaries of participants' pre-existing medical conditions will be presented by MedDRA SOC, PT, and Dose Cohort (Table 14).

Individual participant listings will be presented for all medical conditions (Listing 7).

#### 9.1.2. Prior and Concomitant Medications

Summaries of medications that were started prior to dosing and continued at the time of dosing will be presented by WHO Drug Code Level 1, Level 2 and Dose Cohort (Table 76).

Individual participant listings will be presented for all prior concomitant medications (Listing 17).

# **9.2.** Measurements of Treatment Compliance

Any participants who were enrolled but did not receive the infusion of study product will be presented by Dose Cohort as part of the participant disposition table (Table 6). A summarized list of dates of dosing by Dose Cohort and site is presented in Table 8.

Date and time of study product administration, along with information on whether the participant was dosed according to protocol will be included in Listing 8. A listing of infusion interruptions will be presented in Listing 9.

#### 9.3. Adverse Events

A treatment-emergent AE (TEAE) is defined as an AE that occurs during or after the study product infusion and up through the final visit. Only TEAEs will be documented as AEs in this study. When calculating the proportions of participants with AEs within a given MedDRA category, each participant will be counted once and any repetitions of AEs within a participant will be ignored, and the event will be reported according to the highest severity recorded (separately for related and unrelated AEs, when both severity and relatedness are tabulated). The denominators for percent values will be indicated within the table or table header.

An overall summary of AEs by Dose Cohort will be presented in Table 23.

The number of AEs and number and proportion of participants reporting an AE or SAE that occurred in  $\geq$ 5% of participants in any Dose Cohort will be presented by MedDRA SOC, and PT (Table 24).

## 9.3.1. Solicited Events and Symptoms

Solicited AEs will be collected from the end of the infusion through Day 3. Solicited AEs will be summarized by severity for each day post administration (Days 1-3) and as the maximum severity over all 3 days. Additionally, solicited AEs will be analyzed using standard techniques, such as exact CIs, to summarize the proportion of participants reporting each symptom. Solicited AEs include headache, rash, nausea, vomiting, diarrhea, fatigue, and myalgia.

The proportion of participants reporting at least one solicited AE will be summarized for each solicited AE. The 95% CI calculated using Clopper-Pearson methodology from a binomial distribution (SAS Proc Freq with a binomial option) will be presented (Table 25).

- The maximum severity of solicited symptoms per participant by day will be presented graphically in Figure 3.
- The proportion of participants experiencing solicited events, Clopper-Pearson 95% CI, and difference of proportion from the placebo group will be summarized in Table 26.
- The number and percentage of participants experiencing solicited events by symptom, maximum severity, will be summarized in Table 27.
- The number and percentage of participants experiencing solicited events by symptom, maximum severity and day after infusion will be summarized in Table 28, Table 29, Table 30, and Table 31.
- Solicited AEs by participant will be presented in Listing 11.

#### 9.3.2. Unsolicited Adverse Events

Unsolicited AEs will be collected from the time of infusion through Day 29. Unsolicited AEs will be coded by MedDRA for PT, HLGT, and SOC. The proportion of participants reporting at least one unsolicited AE will be summarized by MedDRA SOC, HLGT and PT post infusion. Denominators for percentages are the number of participants who received the infusion being summarized.

AEs by participant will be presented in Listing 12.

The following summaries for unsolicited AEs will be presented by MedDRA SOC, HLGT, PT, and Dose Cohort:

- The incidence and total frequency of AEs with Pearson-clopper 95% CI (Table 32)
- Summary of maximum severity and relationship to study product (Table 33 and Table 34)
- Participant incidence and total frequency of related adverse events by Dose Cohort (Table 35)
- Participant listing of serious AEs (Table 36)
- Participant listing of non-serious AEs of moderate or severe grade (Table 37)
- Listing of other significant AEs (Table 38)
- Listing of Unanticipated Problems (UPs) (Table 39, Table 40)
- Bar chart of non-serious related AEs by severity and MedDRA SOC (Figure 4)
- Bar chart of non-serious related AEs by maximum severity and MedDRA SOC (Figure 5)

# 9.4. Deaths, Serious Adverse Events and other Significant Adverse Events

The following listings will be presented including Participant ID, Age (years), Adverse Event Description, Adverse Event Onset Date/End Date, Dose Received/Days Post Dose, Reason Reported as an SAE, Relationship to Treatment, Alternate Etiology if not Related, Outcome, and Duration of Event (days):

- Deaths and Serious Adverse Events (Table 36)
- Non-serious unsolicited, moderate or severe AEs, which are grade 2 or more (Table 37)

Other significant AEs, including NOCMCs, MAAEs, (Table 38) and UPs (Table 39, Table 40).

## 9.5. Pregnancies

For any participants in the Safety Population who became pregnant during the study, every attempt will be made to follow these participants to completion of pregnancy to document the outcome, including information regarding any complications with pregnancy and/or delivery. Listings of pregnancies and outcomes will be presented (Listing 19, Listing 20, Listing 21, Listing 22, and Listing 23).

# 9.6. Clinical Laboratory Evaluations

Clinical evaluations will be done to evaluate safety endpoints. These evaluations will include monitoring and recording of AEs and SAEs, clinical safety laboratory test results, VS measurements, 12-lead ECG results, and physical examination findings. The timing and frequency of all safety assessments are listed in the SOA (Table 2).

Toxicity grading criteria for clinical laboratory results can be found in Table 5. Unscheduled clinical laboratory evaluations will be included in listings but excluded from tabular and graphical summaries, except when calculating the maximum severity post-baseline. Any pre-existing abnormal lab results at Screening and Baseline will be graded and presented in listings. The following parameters will be presented (in order): Chemistry - Creatinine, Total Bilirubin, ALT; Hematology - Hemoglobin (Hgb), WBC, Platelets (PLT); Hypersensitivity testing. Hypersensitivity testing will be conducted if a participant experiences anaphylaxis or an anaphylactoid event related to the infusion. One sample will be obtained at approximately 15 minutes prior to the infusion; if the participant experiences a reaction, three additional samples will be drawn: 1) at the onset of symptoms, 2) 2 or more hours after onset of symptoms, and 3) after resolution of symptoms. The hypersensitivity panel will measure complement levels and activity (C3, C4, and CH50), Immunoglobulin E (IgE) levels, and tryptase on serum.

Participants with abnormal laboratory results, which are Grade 1 or higher, will be listed in Table 41, Table 42, and Table 43 for chemistry, hematology, and hypersensitivity, respectively. A full listing with all laboratory results will be listed in Listing 1 and Listing 2 for chemistry and hematology, respectively.

#### 9.6.1. Clinical Laboratory Evaluations – Chemistry

Summaries of the number of participants with chemistry laboratory results, by grade severity, will be presented in Table 44, Table 45, Table 46, and Table 47.

Summaries of the number of participants with abnormal chemistry laboratory results related to study treatment, by grade severity, will be presented in Table 48, Table 49, Table 50, and Table 51.

Descriptive statistics including mean, SD, median, minimum and maximum values by time point, and changes from baseline, for each laboratory parameter will be summarized in Table 52, Table 53, and Table 54.

Changes in laboratory values will be presented in Figure 6, Figure 7, and Figure 8 for Creatinine, Total Bilirubin, and ALT, respectively.

#### 9.6.2. Clinical Laboratory Evaluations - Hematology

A summary of the number of participants with hematology laboratory results, by grade severity, will be presented in Table 55, Table 56, Table 57, Table 58 and Table 59.

A summary of the number of participants with abnormal hematology laboratory results related to study treatment, by grade severity, will be presented in Table 60, Table 61, Table 62, Table 63, and Table 64.

Descriptive statistics including mean, SD, median, minimum and maximum values by time point, and changes from baseline, for each hematology laboratory parameter, will be summarized in Table 65, Table 66, and Table 67. Changes in laboratory values will be presented in Figure 9, Figure 10, and Figure 11 for Hgb, WBC, and PLT, respectively.

# 9.7. Vital Signs and Physical Examinations

Toxicity grading criteria for VS results can be found in Table 5. Vital signs will be obtained on Day 1, Day 2, Day 3, Day 8, Day 15, and Day 29 of the study. Unscheduled VS measurements will be listed, but excluded from tabular and graphical summaries by time point, except when calculating the maximum severity post baseline. Refer to Section 3.3.1 for the definition of baseline. If VS measurements are repeated, the following rules will be used to determine which VS measurement to use for analyses if repeat measurements occur:

- 1. If the first replicate is normal, then it will be used for analysis.
- 2. If the first and second replicates are both abnormal, then the replicate with the higher severity will be used for analysis.
- 3. If the first replicate is abnormal, the second replicate is normal, and the third replicate was not performed, then the first replicate will be used in the analysis.
- 4. If the first replicate is abnormal, the second replicate is normal, and the third replicate is normal, then the second replicate will be used in the analysis.
- 5. If the first replicate is abnormal, the second replicate is normal, and the third replicate is abnormal, then the abnormal replicate with the higher severity will be used for analysis.

VS parameters that have grading criteria for both decreases (result lower than normal range) and increases (result higher than normal range) will be summarized separately by direction.

VS results will be summarized in tables by parameter, Dose Cohort, and time point (Table 68, Table 69, Table 70, Table 71, Table 72, Table 73, and Table 74.

All individual VS measurements, including height, weight, and oximetry measurements (SpO<sub>2</sub>) will be presented in Listing 15.

Focused physical examinations performed on Day 1, Day 3, and Day 8. Symptom-driven physical examinations performed on Day 15, Day 29, Day 61, Day 91 and Day 121 if indicated based on review of complete medical history and any updates obtained by interview of participants since the previous visit.

Abnormal physical exam findings will be presented in Listing 16.

# 9.8. 12-Lead Standard Electrocardiogram

Summary of 12-lead standard ECG change in overall interpretation from baseline will be shown by Dose Cohort and time point (Table 75).

A listing of ECG overall interpretations and comments will be presented in Listing 24.

#### 9.9. Prior and Concomitant Medications

Prior and concomitant medications will be coded to the Anatomical Therapeutic Classification using the WHO Drug Dictionary. The use of prior and concomitant medications taken during the study will be recorded on the CRFs. A by-participant listing of concomitant medication use will be presented. The use of concomitant medications during the study will be summarized by WHO Drug Code Level 1, Level 2 and Dose Cohort (Table 76). Individual participant listings will be presented for all prior concomitant medications (Listing 17).

# 9.10. Other Safety Measures

Not Applicable.

#### 10. PHARMACOKINETICS

EV68-228-N concentrations and PK parameters will be summarized by Dose Cohort. Statistics include the arithmetic mean, median, SD, geometric mean (GM), coefficient of variation (CV), minimum, and maximum. CV will be calculated using the method for log-normally distributed data and reported as a percent:

 $CV\% = \sqrt{\exp(s^2) - 1} \times 100\%$ , where s<sup>2</sup> is the standard deviation of the log-transformed data

# 10.1. Summary of Pharmacokinetic Sampling and Sample Properties

The serum PK of a single dose of EV68-228-N will be assessed from serial blood samples collected approximately 15 minutes prior to infusion, at end of infusion (within a  $\pm$  5-minute window), at 1-, 3-, and 5-hours post end of infusion (within a  $\pm$  15-minute window), at 24- and 48-hours after the end of the infusion (within  $\pm$ 3-hour window), and at 7, 14, 28, 60, 90, and 121 days after the end of the infusion (within  $\pm$ 1-, 2-, 3-, 7-, 14-, and 14-day window, respectively). EV68-228-N will be quantified by a validated ECL assay.

Individual concentration-time plots will be generated, and outliers will be identified as values greater or less than 3 SDs from the mean within each Dose Cohort and time point. Outliers will not be excluded from summary statistics but will be excluded from the NCA and will be discussed in the CSR.

Samples with bioanalytical errors or quality issues reported by the laboratory will be excluded. Collection times of samples missing the actual collection time will be imputed using the nominal collection time. Such samples will be identified in the analysis report (Listing 25).

# 10.2. Pharmacokinetic Analysis

#### 10.2.1. Concentration Summaries

EV68-228-N serum concentrations will be listed by Dose Cohort and participant. Out-of-window sample time and PK analyses-excluded samples will be indicated, as will BQL values that were imputed for the purposes of parameter estimation (Listing 25). The listings will also indicate the nominal and actual time associated with the sample (nominal time is defined as the planned time in minutes, hours, or days since the first dose). Potentially important bioanalytical errors and their effect on the PK analysis will be discussed.

Concentrations below the quantitation limit (BQL) prior to the first measurable concentration will be imputed as zero. The first BQL concentration reported in the serum concentrations after the last measurable concentration may be imputed for the purpose of parameter estimation as the LLOQ divided by 2 only if 1) needed to estimate  $\lambda z$ , 2) all other  $\lambda z$  estimation criteria are met, and 3) if a visual predictive check of the imputed value appears to be consistent with the observed elimination trend. All other BQL samples will be treated as missing. Imputed concentration values will only be used for serum parameter estimation by NCA and not included in concentration summaries, however, imputed BQL values will be indicated by imputation method in listings with methods clarified in the footnote and denoted in figures.

EV68-228-N serum concentrations will also be summarized by Dose Cohort (Table 77 and Table 78) and plotted by Dose Cohort. Figure 12, Figure 13, and Figure 14 will present the participant serum concentration profiles using a linear plot and Figure 15, Figure 16, and Figure 17 will present the participant serum concentration using a semilogarithmic plot. Linear plots of serum mean concentration curves will be shown in Figure 18, with error bars representing ± 1 SD. Semi-logarithmic plots of geometric mean serum concentration curves will be shown in Figure 19.

#### 10.2.2. Pharmacokinetic Parameters

PK analyses will be performed using noncompartmental analysis (NCA) using Phoenix WinNonlin version 8.3 or higher (Certara, Radnor, PA).

NCA PK parameters will be calculated using the actual post-dose time. Samples with concentrations greater than the LLOQ will be considered for the estimation of  $\lambda z$ . Imputing the first BQL concentration following the last concentration greater than LLOQ to LLOQ divided by 2 will be considered on a participant-by-participant basis for participants where the  $\lambda z$  acceptance criteria are not met by the observed data greater than the LLOQ.  $\lambda z$  will be computed from the log-transformed concentration data. The correlation between time and concentration at the time points used to estimate  $\lambda z$  should be sufficiently high (adjusted-R<sup>2</sup> >0.9). Additionally, a minimum of three concentrations in the terminal elimination phase will be used for the calculation of  $\lambda z$ . All concentrations used to calculate  $\lambda z$  must come from samples taken at or after  $T_{max}$ . The concentrations used to calculate  $\lambda z$  along with the number of concentrations used for the calculation will be included in the participant serum concentration listing (Listing 25).

The serum AUC will be computed using the linear-up log-down (linear-log) trapezoidal method.

All serum PK parameters will also be summarized by Dose Cohort using descriptive statistics (Table 80). Additionally, participant-level PK parameters will be presented by participant in Table 79 in the final report.

The following parameters will be estimated:  $AUC_{0-\infty}$ ,  $AUC_{0-last}$ ,  $AUC_{0-48}$ ,  $C_{max}$ ,  $T_{max}$ ,  $t_{1/2}$ , CL, and  $V_z$ . See Section 3.3.4 for parameter definitions.

#### 11. IMMUNOGENICITY

The immunogenicity data, determined by a validated ADA assay (14), will be analyzed with mITT and Per-Protocol populations. The proportion of participants with positive screening assay results and positive confirmation assay results are summarized in Table 15, Table 16, Table 17, and Table 18.

A titer assay will be performed for specimens with detectable ADA (refer to Section 3.3.3 for the definition of detectable ADA). Geometric Mean Titers (GMT) of ADAs will be calculated, along with 95% CIs, for all groups, at each time point (Table 19 and Table 20). Summaries will also be displayed graphically (Figure 2).

The GMT is defined as:

$$GMT = \sqrt[n]{X_1 * X_2 * \dots * X_n},$$

where the  $X_1, X_2, ... X_n$  are the titers for each participant at a certain time point for detectable ADAs. In practice, it is the equivalent of:  $GMT = Exp\{[log(X_1) + log(X_2) + ... + log(X_n)] / n\}$ 

The proportion of participants with detectable ADAs and Clopper-Pearson exact 95% CIs will also be computed over time to assess persistence of ADAs (Table 21 and Table 22).

The individual ADA results, including screening result, confirmatory result and titers, will be presented in Listing 10.
#### **12. OTHER ANALYSES**

Not Applicable.

#### 13. REPORTING CONVENTIONS

The mean, SD, and other statistics will be reported to 1 decimal place greater than the original data. The minimum and maximum will use the same number of decimal places as the original data. Proportions will be presented as 2 decimal places; values greater than zero but <0.01 will be presented as "<0.01". Percentages will be reported to the nearest whole number; values greater than zero but < 1% will be presented as "<1"; values greater than 99% but less than 100% will be reported as >99%.

Drug concentrations, AUC values,  $C_{max}$  and their summary statistics will have the same format as the drug concentrations reported by the bioanalytical laboratory. Other PK parameters will be reported to 1 decimal place.

## 14. TECHNICAL DETAILS

SAS version 9.4 or above will be used to generate all tables, figures and listings.

# 15. SUMMARY OF CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSES

Not applicable.

#### 16. REFERENCES

- 1. Murphy OC, Messacar K, Benson L, Bove R, Carpenter JL, Crawford T, et al. Acute flaccid myelitis: cause, diagnosis, and management. Lancet. 2021;397(10271):334-46.
- 2. Marchese DL, Feldman K, Sinn C, Javaid S, Jaffe A, Katz E, et al. Rehabilitation Outcomes in Children With Acute Flaccid Myelitis From 2014 to 2019: A Multicenter Retrospective Review. Pediatr Neurol. 2023;145:41-7.
- 3. Messacar K, Schreiner TL, Van Haren K, Yang M, Glaser CA, Tyler KL, et al. Acute flaccid myelitis: A clinical review of US cases 2012-2015. Ann Neurol. 2016;80(3):326-38.
- 4. Vogt MR, Wright PF, Hickey WF, De Buysscher T, Boyd KL, Crowe JE, Jr. Enterovirus D68 in the Anterior Horn Cells of a Child with Acute Flaccid Myelitis. N Engl J Med. 2022;386(21):2059-60.
- 5. Centers for Disease Control and Prevention. AFM Cases and Outbreaks: CDC; 2023 [updated 04 APR 2023; cited 2023. Available from: https://www.cdc.gov/acute-flaccid-myelitis/cases-in-us.html.
- 6. Vogt MR, Fu J, Kose N, Williamson LE, Bombardi R, Setliff I, et al. Erratum for Research Article "Human antibodies neutralize enterovirus D68 and protect against infection and paralytic disease," by Matthew R. Vogt, Jianing Fu, Nurgun Kose, Lauren E. Williamson, Robin Bombardi, Ian Setliff, Ivelin S. Georgiev, Thomas Klose, Michael G. Rossmann, Yury A. Bochkov, James E. Gern, Richard J. Kuhn, James E. Crowe Jr. Sci Immunol. 2020;5(51).
- 7. KBio Inc. EV68-228-N Investigator's Brochure. 2022.
- 8. Malik P, Edginton A. Pediatric physiology in relation to the pharmacokinetics of monoclonal antibodies. Expert Opin Drug Metab Toxicol. 2018;14(6):585-99.
- 9. Temrikar ZH, Suryawanshi S, Meibohm B. Pharmacokinetics and Clinical Pharmacology of Monoclonal Antibodies in Pediatric Patients. Paediatr Drugs. 2020;22(2):199-216.
- 10. Jacob S NA, Morsy MA. Dose conversion between animals and humans: A practical solution. Indian Journal of Pharmaceutical Education and Research. 2022;56(3):7.
- 11. U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER). Guidance for Industry: Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers. Rockville, MD: Center for Drug Evaluation and Research (CDER); July 2005. p. 27.
- 12. Iwasaki A. Immune Regulation of Antibody Access to Neuronal Tissues. Trends Mol Med. 2017;23(3):227-45.
- 13. U.S. Department of Health and Human Services. Common Terminology Criteria for Adverse Events (CTCAE) 2017 [cited 2023 13 APR]. Available from: <a href="https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/ctcae\_v5\_quick\_reference\_5x7.pdf">https://ctep.cancer.gov/protocoldevelopment/electronic\_applications/docs/ctcae\_v5\_quick\_reference\_5x7.pdf</a>.
- 14. U.S. Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER), Center for Biologics Evaluation and Research (CBER). Guidance for Industry: Immunogenicity Testing of Therapeutic Protein Products Developing and Validating Assays for
- 15. Anti-Drug Antibody Detection. January 2019.

## 17. LISTING OF TABLES, FIGURES, AND LISTINGS

Table, figure, and listing shells are presented in Appendices 1, 2, and 3.

# **APPENDICES**

| <b>APPENI</b> | DIX 1. TABLE MOCK-UPS | |
|---|---|---|
| Table 1: | Single Ascending Dose Cohorts and Dose Regimens | 48 |
| Table 2: | Schedule of Activities | 49 |
| Table 3: | Probability to Observe at Least n AEs Within Study Population | 51 |
| Table 4: | Distribution of Protocol Deviations by Category, Type, and Dose Cohort – All Enrolled Participants. | 52 |
| Table 5: | Laboratory Adverse Event Grading Scale | 54 |
| Table 6: | Participant Disposition by Dose Cohort – All Enrolled Participants | 55 |
| Table 7: | Analysis Populations by Dose Cohort – All Enrolled Participants | 56 |
| Table 8: | Dates of Treatment by Site and Dose Cohort | 57 |
| Table 9: | Ineligibility Summary of Screen Failures | 58 |
| Table 10: | Summary of Categorical Demographic and Baseline Characteristics by Site | 59 |
| Table 11: | Summary of Continuous Demographic and Baseline Characteristics by Site | 60 |
| Table 12: | Summary of Categorical Demographic and Baseline Characteristics by Dose<br>Cohort – All Enrolled Participants | 61 |
| Table 13: | Summary of Continuous Demographic and Baseline Characteristics by Dose<br>Cohort – All Enrolled Participants | 62 |
| Table 14: | Summary of Participants with Pre-Existing Medical Conditions by MedDRA System Organ Class, Preferred Term and Dose Cohort | 63 |
| Table 15: | Proportion of Participants with a Positive Screening Assay by Time Point and Dose Cohort – mITT Population. | 64 |
| Table 16: | Proportion of Participants with a Positive Screening Assay by Time Point and Dose Cohort – Per-Protocol Population | 64 |
| Table 17: | Summary of Positive ADA Confirmation Assay Results by Time Point and Dose Cohort – mITT Population | 65 |
| Table 18: | Summary of Positive ADA Confirmation Assay Results by Time Point and Dose Cohort – Per-Protocol Population | 65 |
| Table 19: | Anti-Drug Antibodies (ADA) Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Dose Cohort – mITT Population | 66 |
| Table 20: | Anti-Drug Antibodies (ADA) Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Dose Cohort – Per-Protocol Population | 67 |
| Table 21: | Proportion of Participants with Detectable Anti-Drug Antibodies (ADA) with 95% Confidence Intervals by Time Point and Dose Cohort – mITT Population | 68 |

| Table 22: | Proportion of Participants with Detectable Anti-Drug Antibodies (ADA) with 95% Confidence Intervals by Time Point and Dose Cohort – Per-Protocol Population | 69 |
|---|---|---|
| Table 23: | Overall Summary of Adverse Events | 70 |
| Table 24: | Adverse Events Occurring in ≥ 5% of Participants in Any Dose Cohort by MedDRA System Organ Class and Preferred Term and Dose Cohort | 71 |
| Table 25: | Number and Percentage of Participants Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Dose Cohort | 72 |
| Table 26: | Comparison of the Proportion of Participants Experiencing Solicited Events by Dose Cohort | 73 |
| Table 27: | Number and Percentage of Participants Experiencing Solicited Events by Symptom, Maximum Severity, and Dose Cohort | 74 |
| Table 28: | Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – 3 mg/kg EV68-228-N | 76 |
| Table 29: | Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – 10 mg/kg EV68-228-N | 77 |
| Table 30: | Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – 30 mg/kg EV68-228-N | 77 |
| Table 31: | Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – Placebo | 77 |
| Table 32: | Summary of Unsolicited Adverse Events by MedDRA System Organ Class,<br>High Level Group Term and Preferred Term and Dose Cohort | 78 |
| Table 33: | Unsolicited Adverse Events by MedDRA System Organ Class, High Level Group Term and Preferred Term, Maximum Severity, and Dose Cohort | 79 |
| Table 34: | Unsolicited Adverse Events by MedDRA System Organ Class, High Level Group Term and Preferred Term, Maximum Severity, Relationship, and Dose Cohort | 80 |
| Table 35: | Related Unsolicited Adverse Events Post Dosing by MedDRA System<br>Organ Class, High Level Group Term and Preferred Term, and Dose Cohort | 82 |
| Table 36: | Listing of Serious Adverse Events | 83 |
| Table 37: | Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events | 84 |
| Table 38: | Listing of Other Significant Adverse Events | 85 |
| Table 39: | Listing of Participant-Specific Unanticipated Problems (UPs) | 86 |
| Table 40: | Listing of Non-Participant Specific Unanticipated Problems (UPs) | 87 |
| Table 41: | Listing of Abnormal Laboratory Results – Chemistry | 89 |
| Table 42: | Listing of Abnormal Laboratory Results – Hematology | 90 |
| Table 43: | Listing of Abnormal Laboratory Results – Hypersensitivity | 91 |

| Table 44: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Chemistry Parameter | 92 |
|---|---|---|
| Table 45: | Laboratory Results by Parameter Time Point, and Dose Cohort – Chemistry: Creatinine | 94 |
| Table 46: | Laboratory Results by Parameter Time Point, and Dose Cohort – Total Bilirubin | 95 |
| Table 47: | Laboratory Results by Parameter Time Point, and Dose Cohort – ALT | 95 |
| Table 48: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Chemistry Parameter | 96 |
| Table 49: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Creatinine | 97 |
| Table 50: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Total Bilirubin | 97 |
| Table 51: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – ALT | 97 |
| Table 52: | Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort - Creatinine | 98 |
| Table 53: | Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – Total Bilirubin | 99 |
| Table 54: | Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort - ALT | 99 |
| Table 55: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Hematology Parameter | 100 |
| Table 56: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – Hemoglobin | 101 |
| Table 57: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – WBC: Low | 101 |
| Table 58: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – WBC: High | 101 |
| Table 59: | Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – Platelets | 101 |
| Table 60: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Hematology Parameter | 102 |
| Table 61: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Hemoglobin | 103 |
| Table 62: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – WBC – Low | 103 |

| Table 63: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – WBC – High | 103 |
|---|---|---|
| Table 64: | Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Platelets | 103 |
| Table 65: | Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort - Hemoglobin | 104 |
| Table 66: | Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort - WBC | 105 |
| Table 67: | Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – Platelets | 105 |
| Table 68: | Vital Signs by Maximum Severity, Time Point, and Dose Cohort – Any Assessment | 106 |
| Table 69: | Vital Signs by Assessment, Maximum Severity, Time Point, and Dose<br>Cohort – Body Temperature | 107 |
| Table 70: | Vital Signs by Assessment, Maximum Severity, Time Point, and Dose<br>Cohort – Pulse: High | 107 |
| Table 71: | Vital Signs by Assessment, Maximum Severity, Time Point, and Dose<br>Cohort – Pulse: Low | 107 |
| Table 72: | Vital Signs by Assessment, Maximum Severity, Time Point, and Dose<br>Cohort – Systolic Blood Pressure: High | 107 |
| Table 73: | Vital Signs by Assessment, Maximum Severity, Time Point, and Dose<br>Cohort – Systolic Blood Pressure: Low | 107 |
| Table 74: | Vital Signs by Assessment, Maximum Severity, Time Point, and Dose<br>Cohort – Diastolic Blood Pressure: High | 107 |
| Table 75: | Summary of Post Dose ECG Change in Overall Interpretations from Baseline by Dose Cohort and Time Point | 108 |
| Table 76: | Number and Percentage of Participants with Prior and Concurrent<br>Medications by WHO Drug Classification and Dose Cohort | 109 |
| Table 77: | Individual Statistics of Serum EV68-228-N Concentrations by Time Point | 110 |
| Table 78: | Summary Statistics of Serum EV68-228-N Concentrations by Time Point | 111 |
| Table 79: | Individual Statistics of Noncompartmental Serum PK Parameters by Dose Cohort | 113 |
| Table 80: | Summary Statistics of Noncompartmental Serum PK Parameters by Dose Cohort | 114 |

## 9.1 Overall Study Design and Plan Description

**Table 1:** Single Ascending Dose Cohorts and Dose Regimens

| Cohort | Arm | Number of Participants | Study Product |
|--------|-----|------------------------|------------------------|
| 1 | 1 | 10 | 3 mg/kg of EV68-228-N |
| I | 2 | 2 | Placebo |
| 2 | 1 | 10 | 10 mg/kg of EV68-228-N |
| 2 | 2 | 2 | Placebo |
| 2 | 1 | 10 | 30 mg/kg of EV68-228-N |
| 3 | 2 | 2 | Placebo |

## 9.5.1 Immunogenicity and Safety Measurements Assessed and Flow Chart

**Table 2:** Schedule of Activities

| Study Visit | 00 | 01 | 02 | 03 | 04 | 05 | 06 | 07 | 08 | 09 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study day | -28 to -1 | 1 | 2 | 3 | 8 | 15 | 29 | 61 | 91 | 121 | ] | Early |
| Visit window (± number of days) | | | | | 1 | 2 | 3 | 7 | 14 | 14 | Unscheduled | <b>Termination</b> |
| Procedures | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | |
| Demographic Information | X | | | | | | | | | | | |
| Review Eligibility Criteria | X | X | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | |
| Concomitant Medications | X | X | X | X | X | X | X | | | | Xª | X <sup>a</sup> |
| Infusion | | X | | | | | | | | | | |
| Interim Medical History | | X | X | X | X | X | X | X | X | X | X | X |
| Counsel on avoidance of pregnancy | X | X | | | | | | | | | | |
| Full Physical Examination | X | | | | | | | | | | | |
| Focused Physical Examination | | X | X | X | X | | | | | | X <sup>a</sup> | X <sup>a</sup> |
| Symptom-driven Physical Examination | | | | | | X | X | X | X | X | X | X |
| Vital Signs | X | $X^{b}$ | X | X | X | X | X | | | | Xª | X <sup>a</sup> |
| Oximetry Measurement | | $X^{b}$ | | | | | | | | | | |
| Cardiopulmonary Monitoring | | X <sup>c</sup> | | | | | | | | | | |
| Height and Weight (for BMI calculation) | X | | | | | | | | | | | |
| Weight (for dose calculation) | | X | | | | | | | | | | |
| Hematology <sup>d</sup> | X | Xe | X | X | X | | X | | | | | X <sup>a</sup> |
| Chemistry <sup>d</sup> | X | Xe | X | X | X | | X | | | | | Xa |
| 12-Lead ECG | X | Xf | X | | | | | | | | | |
| Urine Pregnancy Test <sup>g</sup> | X | X | | | | | | | | | | |
| Solicited AEs | | | Days 1-3 | | | | | | | | | |

**Table 2: Schedule of Activities** (continued)

| Study Visit | 00 | 01 | 02 | 03 | 04 | 05 | 06 | 07 | 08 | 09 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study day | -28 to -1 | 1 | 2 | 3 | 8 | 15 | 29 | 61 | 91 | 121 | | Early |
| Visit window (± number of days) | | | | | 1 | 2 | 3 | 7 | 14 | 14 | Unscheduled | <b>Termination</b> |
| Procedures | | | | | | | | | | | | |
| Review e-Memory Aid | | | X | X | X | | | | | | | |
| Unsolicited AEs | | | | Days 1 | -29 | | | | | | | |
| SAEs, MAAEs, and NOCMCs | | Days 1-121 | | | | | | | | | | |
| Update previous AE/SAEs (as needed) | | | X | X | X | X | X | X | X | X | X | X |
| PK samples h | | Xi | $\mathbf{X}^{\mathrm{j}}$ | $\mathbf{X}^{\mathrm{j}}$ | X | X | X | X | X | X | | X |
| Serum samples for ADA (anti-drug antibodies)h | | Xe | | | X | X | X | X | X | X | | X |
| Hypersensitivity Panel Samplek | | X <sup>k</sup> | | | | | | | | | | |
| Total amount of blood collected for visit (mL) | 6 | 41 or 56 <sup>l</sup> | 11 | 11 | 16 | 10 | 16 | 10 | 10 | 10 | 0 | 16 |
| Cumulative blood volume (ml) if there is no hypersensitivity reaction | 6 | 47 | 58 | 69 | 85 | 95 | 111 | 121 | 131 | 141 | | |
| Cumulative blood volume (mL) if there is a hypersensitivity reaction | 6 | 62 | 73 | 84 | 100 | 110 | 126 | 136 | 146 | 156 | | |

<sup>&</sup>lt;sup>a</sup> Conducted if visit occurs within 7 days of infusion.

<sup>&</sup>lt;sup>b</sup> VS will be collected to confirm eligibility prior to randomization and will be repeated, along with oximetry measurements, at approximately 15 minutes prior to infusion, the end of infusion, and at 1-hour post-infusion. For infusions lasting at least 30 minutes, these will also be collected at approximately 15 minutes after the beginning of the infusion.

<sup>&</sup>lt;sup>c</sup> During infusion and up to one-hour post-infusion, continuous cardio-pulmonary monitoring will be conducted to assess for acute changes. If a CS change occurs, the monitoring will be continued until it has resolved and it is deemed safe to discontinue monitoring by the site PI or designee.

d Clinical screening laboratory evaluations will include WBCs, Hgb, PLT, Cr, ALT, and T. Bili. Clinical safety laboratory evaluations obtained on Days 1, 2, 3, 8, and 29 will include WBCs, Hgb, PLTs, Cr, ALT, and T. Bili. Results of laboratory studies collected prior to infusion on Day 1 do not require review prior to infusion; rather, they serve as a baseline assessment for post-infusion safety assessment.

e Day 1 blood draws for ADA, hematology and chemistry should be done at the same time as the first PK blood draw, within 15 minutes prior to the infusion

<sup>&</sup>lt;sup>f</sup> ECGs on Day 1 will occur approximately 15 minutes prior to infusion and 1-hour post-infusion.

g For women of childbearing potential, a urine pregnancy test at screening and on Day 1 with results confirmed as negative prior to infusion.

h If an infusion is terminated early, the remaining Day 1 PK samples will not be drawn and the PK and ADA samples at follow-up visits will not be drawn.

<sup>&</sup>lt;sup>1</sup> PK samples on Day 1 will be obtained approximately 15 minutes prior to infusion, at end of infusion (within a + 5-minute window), and at 1-, 3-, and 5-hours post end of infusion, within a ± 15-minute window. Note, for infusions that last longer than 1-hour due to infusion related events or other disruptions in administration, see MOP for details on updating the PK collection timepoints.

<sup>&</sup>lt;sup>j</sup> PK sample will be collected within ±3-hour window of 24- and 48-hours after the end of infusion

k All participants will have a baseline sample taken for hypersensitivity testing approximately 15 minutes prior to infusion. For any participant that has an anaphylactic or anaphylactoid-type reaction, three additional samples will be taken: 1) at the onset of symptoms, 2) at 2 or more hours after onset, 3) at the resolution of symptoms.

<sup>&</sup>lt;sup>1</sup> Larger amount will be collected only if there is a hypersensitivity reaction.

## 9.7.1 Sample Size

**Table 3:** Probability to Observe at Least n AEs Within Study Population

| Adverse Event | Probability to Observe At Least n AEs | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Probability | n=1 | n=2 | n=3 | n=4 | n=5 | n=6 | n=7 | n=8 | n=9 | n=10 |
| 5% | 40.1% | 8.6% | 1.2% | 0.1% | 0.0% | 0.0% | 0.0% | 0.0% | 0.0% | 0.0% |
| 10% | 65.1% | 26.4% | 7.0% | 1.3% | 0.2% | 0.0% | 0.0% | 0.0% | 0.0% | 0.0% |
| 15% | 80.3% | 45.6% | 18.0% | 5.0% | 1.0% | 0.1% | 0.0% | 0.0% | 0.0% | 0.0% |
| 20% | 89.3% | 62.4% | 32.2% | 12.1% | 3.3% | 0.6% | 0.1% | 0.0% | 0.0% | 0.0% |
| 25% | 94.4% | 75.6% | 47.4% | 22.4% | 7.8% | 2.0% | 0.4% | 0.0% | 0.0% | 0.0% |
| 30% | 97.2% | 85.1% | 61.7% | 35.0% | 15.0% | 4.7% | 1.1% | 0.2% | 0.0% | 0.0% |

#### 10.2 Protocol Deviations

Table 4: Distribution of Protocol Deviations by Category, Type, and Dose Cohort – All Enrolled Participants

[Implementation notes: Only include deviation categories/types that exist in the data, if there are none in some category/type then delete the row.]

| | | 3 mg/kg<br>EV68-228-N<br>(N=X) | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | Placebo<br>(N=X) | | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No. of Pts. | No. of<br>Dev. | No. of Pts. | No. of Dev. | No. of Pts. | No. of<br>Dev. | No. of Pts. | No. of Dev. | No. of Pts. | No. of Dev. |
| Major Deviation | | | | | | - | | | | 1 | |
| Eligibility/Enrollment | Any type | | | | | | | | | | |
| | Did not meet inclusion criterion | х | X | x | X | X | X | x | X | x | X |
| | Met exclusion criterion | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Informed Consent/Assent | Any Type | | | | | | | | | | |
| | ICF not signed prior to study procedures | | | | | | | | | | |
| | Incorrect version of ICF signed Unapproved consent/reconsent informed consent method used | | | | | | | | | | |
| Product administration schedule | Any type | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | |
| | Missed treatment administration | | | | | | | | | | |
| | Delayed treatment administration | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Follow-up visit schedule | Any type | | | | | | | | | | |
| | Out of window visit | | | | | | | | | | |
| | Missed visit/visit not conducted | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Protocol procedure/assessment | Any type | | | | | | | | | | |
| | Required procedure not conducted Required procedure done | | | | | | | | | | |
| | incorrectly | | | | | | | | | | |

Table 4: Distribution of Protocol Deviations by Category, Type, and Dose Cohort (continued)

| | | 3 mg/kg<br>EV68-228-N<br>(N=X) | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | Placebo<br>(N=X) | | All Parti | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Category | Deviation Type | No. of Pts. | No. of<br>Dev. | No. of Pts. | No. of<br>Dev. | No. of Pts. | No. of<br>Dev. | No. of Pts. | No. of<br>Dev. | No. of Pts. | No. of<br>Dev. |
| | Safety Lab not Collected | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Laboratory/Specimen | Any type | | | | | | | | | | |
| | Specimen result not obtained Conduct of Non-Protocol Procedure Specimen Processing not conducted correctly | | | | | | | | | | |
| | Specimen Temperature Excursion | | | | | | | | | | |
| | Other | | | | | | | | | | · |
| Product Storage | Any type Study Product Temperature Excursion | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Safety | Any type | | | | | | | | | | |
| | Safety Lab not Collected | | | | | | | | | | · |
| | Required procedure done incorrectly | | | | | | | | | | |
| | Required procedure not conducted | | | | | | | | | | · |
| | Specimen result not obtained | | | | | | | | | | |
| | Other | | | | | | | | | | |
| Repeat for Minor Deviation | • | | | . " | | · ' | | . " | | | |
| Repeat for All Deviations | | | | | | | | | | | |

Note: N=Number of participants enrolled in each group.

## 12.4.1 Individual Laboratory Measurements and Abnormal Laboratory Values

**Table 5:** Laboratory Adverse Event Grading Scale

| Protocol Assessment | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Hematology | | | | |
| Hemoglobin, Low (male) g/dL | 12.0 - 13.0 | 10.0 - 11.9 | 8.0 - 9.9 | <8.0 |
| Hemoglobin, Low (female) g/dL | 10.5 - 11.5 | 9.0 - 10.4 | 7.5 - 8.9 | <7.5 |
| WBC, Low mm <sup>3</sup> | 2,500 - 2,999 | 1,500 - 2,499 | 1,000 - 1,499 | <1,000 |
| WBC, High mm <sup>3</sup> | 11,600 - 15,000 | 15,001 - 20,000 | 20,001 - 25,000 | >25,000 |
| Platelets (Decrease) mm <sup>3</sup> | 125,000 - 139,000 | 100,000 - 124,000 | 25,000 - 99,000 | <25,000 |
| Chemistry | | | | |
| ALT | 2.0 - 3.5x ULN | >3.5 - 5.0x ULN | >5.0 - 10x ULN | >10x ULN |
| Creatinine | 1.5 - 1.7x ULN | >1.7 - 2.0x ULN | >2.0 - 2.5x ULN | >2.5x ULN or requires dialysis |
| Bilirubin | 1.5 - 2.0x ULN | >2.0 - 3.0x ULN | >3.0 - 5.0x ULN | >5.0x ULN |
| Vital Signs | | | | |
| Hypertension (systolic) mmHg | 141 - 150 | 151 - 155 | >155 | ER visit or hospitalization for management |
| Hypertension (diastolic) mmHg | 91 - 95 | 96 - 100 | >100 | ER visit or hospitalization for management |
| Hypotension (systolic) mmHg | 85-89 | 80-84 | <80 | ER visit or hospitalization for management |
| Bradycardia, baseline>60 bpm | 50 - 54 | 45-49 | <45 | ER visit or hospitalization for management |
| Bradycardia, baseline <60 bpm | 45-50 | 40-44 | <40 | ER visit or hospitalization for management |
| Tachycardia bpm | 101 - 115 | 116 - 130 | >130 | ER visit or hospitalization for management |
| Temperature °C | 38.0 - 38.4 | 38.5 - 38.9 | 39.0 - 40.0 | >40 |

#### 14.1 **Description of Study Participants**

#### 14.1.1 Disposition of Participants

Participant Disposition by Dose Cohort - All Enrolled Participants Table 6:

| Participant | 3 mg/kg<br>EV68-228-N<br>(N=X) | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | Placebo<br>(N=X) | | All Participants (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Disposition | n | % | n | % | n | % | n | % | n | % |
| Screened | | | | | | | | | X | |
| Enrolled/Randomized | Х | 100 | X | 100 | X | 100 | Х | 100 | X | 100 |
| Received Treatment | Х | xx | X | XX | X | XX | Х | XX | X | XX |
| Completed Final Blood Draw for Safety at Study<br>Day 29 | х | xx | X | XX | X | xx | X | XX | X | xx |
| Completed at Least One Post-Dose Blood Draw for PK | х | xx | X | xx | Х | xx | х | XX | х | xx |
| Completed Final Blood Draw for ADA at Study Day 121 | х | xx | x | xx | х | xx | х | XX | х | xx |
| Terminated from the study follow-up | X | xx | Х | XX | X | XX | Х | xx | X | XX |
| Completed Follow-up (Study Day 121) <sup>a</sup> | X | xx | х | XX | X | xx | Х | XX | X | XX |
| Completed Per Protocol <sup>b</sup> | Х | xx | X | XX | X | XX | X | XX | X | XX |

Note: N=Number of participants enrolled in each group.

a Refer to Listing 16.2.1 for reasons participants discontinued or terminated early.

b Refer to Listing 16.2.3 for reasons participants are excluded from the Analysis populations.

**Table 7:** Analysis Populations by Dose Cohort – All Enrolled Participants

| Analysis | | 3 mg/kg<br>EV68-228-N<br>(N=X) | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | Placebo<br>(N=X) | | All Participants (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Populations | Reason Participants Excluded | n | % | n | % | n | % | n | % | % | n |
| Safety | Any Reason | х | XX | Х | XX | X | XX | X | XX | Х | XX |
| Population | [Reason 1, for example: Did not receive study product] | | | | | | | | | | |
| mITT Population | Any Reason | | | | | | | | | | |
| | Did not receive at least a partial study product | | | | | | | | | | |
| | Did not have a valid pre-dose immunogenicity testing result | | | | | | | | | | |
| | Did not have any valid post-dose immunogenicity testing result | | | | | | | | | | |
| Per-Protocol | Any Reason | | | | | | | | | | |
| Population | Excluded from mITT | | | | | | | | | | |
| | Found to be ineligible at baseline. | | | | | | | | | | |
| | [Reason 3] | | | | | | | | | | |
| | [Reason 4] | | | | | | | | | | |
| Pharmacokinetics | Any Reason | | | | | | | | | | |
| Population | Did not receive a full dose of study product. | | | | | | | | | | |
| | Do not have at least one evaluable serum PK samples for the estimation of $C_{max}$ OR $AUC_{0-\infty}$ | | | | | | | | | | |
| | [Reason 3] | | | | | | | | | | |
| | [Reason 4] | | | | | | | | | | |

Note: N=Number of participants enrolled in each group.

**Table 8:** Dates of Treatment by Site and Dose Cohort

[Implementation Note: The dates of dosing will be categorized by 3 months period (from first enrollment in each cohort).]

| Dates of Dosing | University of<br>Maryland<br>EV68-228-N<br>(N=X) | University of<br>Maryland<br>Placebo<br>(N=X) | Vanderbilt<br>University<br>EV68-228-N<br>(N=X) | Vanderbilt<br>University<br>Placebo<br>(N=X) | All Sites<br>EV68-228-N<br>(N=X) | All Sites<br>Placebo<br>(N=X) | All Sites All Participants (N=X) |
|---|---|---|---|---|---|---|---|
| Total (Entire period of enrollment) | | | | | | | |
| | • | Cohort 1 | | • | | | |
| DDMMMYYYY-DDMMMYYYY [categorize based on length of enrollment period] | X | x | x | x | x | X | х |
| | | Cohort 2 | | | | | |
| DDMMMYYYY-DDMMMYYYY [categorize based on length of enrollment period] | x | x | x | x | x | х | x |
| | | Cohort 3 | | | | | |
| DDMMMYYYY-DDMMMYYYY [categorize based on length of enrollment period] | x | x | x | x | x | x | x |

Note: N=Number of participants enrolled in each group.

Table 9: **Ineligibility Summary of Screen Failures** 

| Inclusion/Exclusion Category | Inclusion/Exclusion Criterion | n <sup>a</sup> | % b |
|---|---|---|---|
| Inclusion and Exclusion | Number of participants failing any eligibility criterion | X | 100 |
| Inclusion | Any inclusion criterion | X | XX |
| | [inclusion criterion 1] | X | XX |
| | [inclusion criterion 2] | X | XX |
| | [inclusion criterion 3] | X | XX |
| Exclusion | Any exclusion criterion | X | XX |
| | [exclusion criterion 1] | X | XX |
| | [exclusion criterion 2] | X | XX |
| | [exclusion criterion 3] | X | XX |
| Eligible but not enrolled | | X | - |

<sup>&</sup>lt;sup>a</sup> More than one criterion may be marked per participant.
<sup>b</sup> Denominator for percentages is the total number of screen failures.

# 14.1.2 Demographic Data by Study Group

Table 10: Summary of Categorical Demographic and Baseline Characteristics by Site

| | | | University of Maryland (N=X) | | University<br>X) | All Parti | |
|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % |
| Sex | Male | х | xx | X | xx | X | XX |
| | Female | | | | | | |
| Ethnicity | Not Hispanic or Latino | X | xx | X | xx | X | XX |
| | Hispanic or Latino | | | | | | |
| | Not Reported | | | | | | |
| | Unknown | | | | | | |
| Race | American Indian or Alaska Native | x | xx | X | xx | X | XX |
| | Asian | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | |
| | Black or African American | | | | | | |
| | White | | | | | | |
| | Multi-Racial | | | | | | |
| | Unknown | | | | | | |

Note: N=Number of participants enrolled in each site.

Table 11: Summary of Continuous Demographic and Baseline Characteristics by Site

| Variable | Statistic | University of Maryland (N=X) | Vanderbilt University (N=X) | All Participants<br>(N=X) |
|---|---|---|---|---|
| Age (yrs) | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (min, max) | xx.x (x.x, x.x) | xx.x (x.x, x.x) | xx.x (x.x, x.x) |
| Height (cm) | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (min, max) | xx.x (x.x, x.x) | xx.x (x.x, x.x) | xx.x (x.x, x.x) |
| Weight (kg) | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| | Median (min, max) | xx.x (x.x, x.x) | xx.x (x.x, x.x) | xx.x (x.x, x.x) |
| BMI (kg/m <sup>2</sup> ) | Mean (SD) | xx.x (xx.x) | xx.x (xx.x) | xx.x (xx.x) |
| , - , | Median (min, max) | xx.x (x.x, x.x) | xx.x (x.x, x.x) | xx.x (x.x, x.x) |

Notes: N=Number of participants enrolled in each site.

BMI is calculated with the height obtained at screening and the weight obtained at Day 1 prior dosing.

Table 12: Summary of Categorical Demographic and Baseline Characteristics by Dose Cohort – All Enrolled Participants

| | | 3 mg/kg<br>EV68-228-N<br>(N=X) | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | Placebo<br>(N=X) | | All Participants (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Variable | Characteristic | n | % | n | % | n | % | n | % | n | % |
| Sex | Male | Х | XX | X | XX | х | XX | X | XX | X | XX |
| | Female | | | | | | | | | | |
| Ethnicity | Not Hispanic or Latino | Х | XX | X | XX | X | XX | x | XX | х | XX |
| | Hispanic or Latino | | | | | | | | | | |
| | Not Reported | | | | | | | | | | |
| | Unknown | | | | | | | | | | |
| Race | American Indian or Alaska Native | х | XX | х | XX | х | XX | x | XX | х | xx |
| | Asian | | | | | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | | | | | |
| | Black or African American | | | | | | | | | | |
| | White | | | | | | | | | | |
| | Multi-Racial | | | | | | | | | | |
| | Unknown | | | | | | | | | | |

Note: N=Number of participants enrolled in each group.

**Summary of Continuous Demographic and Baseline Characteristics by Dose Cohort – Table 13: All Enrolled Participants** 

| Variable | Statistic | 3 mg/kg<br>EV68-228-N<br>(N=X) | 10 mg/kg<br>EV68-228-N<br>(N=X) | 30 mg/kg<br>EV68-228-N<br>(N=X) | Placebo<br>(N=X) | All Participants<br>(N=X) |
|---|---|---|---|---|---|---|
| Age (yrs) | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median (min, max) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) | xx.x (xx.x,<br>xx.x) | xx.x (xx.x, xx.x) |
| Height (cm) | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median (min, max) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| Weight (kg) | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median (min. max) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |
| BMI (kg/m2) | Mean (SD) | xx (xx) | xx (xx) | xx (xx) | xx (xx) | xx (xx) |
| | Median (min, max) | x (x, x) | x (x, x) | x (x, x) | x (x, x) | x (x, x) |

Notes: N=Number of participants enrolled in each group.

BMI is calculated with the height obtained at screening and the weight obtained at Day 1 prior dosing.

### 14.1.3 Prior and Concurrent Medical Conditions

Table 14: Summary of Participants with Pre-Existing Medical Conditions by MedDRA System Organ Class, Preferred Term and Dose Cohort

| MedDRA System | MedDRA Preferred - | 3 mg/kg<br>EV68-228-N<br>(N=X) | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | Placebo<br>(N=X) | | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Organ Class | Term | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any PT | X | XX | X | XX | X | XX | X | XX | x | XX |
| [SOC 1] | Any PT | | | | | | | | | | |
| | PT1 | | | | | | | | | | |
| | PT2 | | | | | | | | | | |
| [SOC 2] | Any PT | | | | | | | | | | |
| | PT1 | | | | | | | | | | |
| | PT2 | | | | | | | | | | |

Notes: N=Number of participants enrolled in each group; n=Number of participants reporting medical history within the specified SOC and PT. A participant is only counted once per SOC and per PT.

### 14.2 Immunogenicity Data

Table 15: Proportion of Participants with a Positive Screening Assay by Time Point and Dose Cohort – mITT Population

| | EV68- | g/kg<br>-228-N<br>=X) | EV68- | ng/kg<br>-228-N<br>=X) | EV68- | ng/kg<br>-228-N<br>=X) | Placebo<br>(N=X) | | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | n | % | n | % | n | % | n | % | n | % |
| Day 1, Pre Dose | X | xx | X | xx | X | XX | X | XX | X | XX |
| Day 8 | | | | | | | | | | |
| Day 15 | | | | | | | | | | |
| Day 29 | | | | | | | | | | |
| Day 61 | | | | | | | | | | |
| Day 91 | | | | | | | | | | |
| Day 121 | | | | | | | | | | |

Note: N=Number of participants in each group in the mITT Population.

Table with similar format:

Table 16: Proportion of Participants with a Positive Screening Assay by Time Point and Dose Cohort – Per-Protocol Population

# Table 17: Summary of Positive ADA Confirmation Assay Results by Time Point and Dose Cohort – mITT Population

[Implementation note, if there is number of participants with positive Screening result is N=0, then the cell will be '-'.]

| | 3 mg/kg<br>EV68-228-N | 10 mg/kg<br>EV68-228-N | 30 mg/kg<br>EV68-228-N | Placebo | All Participants |
|---|---|---|---|---|---|
| Time Point | n/N | n/N | n/N | n/N | n/N |
| Day 1, Pre Dose | x/X | x/X | x/X | x/X | x/X |
| Day 8 | | | | | |
| Day 15 | | | | | |
| Day 29 | | | | | |
| Day 61 | | | | | |
| Day 91 | | | | | |
| Day 121 | | | | | |

Notes: N=Number of participants with positive screening results in each group in the mITT Population. n=Number of participants with positive confirmation results in each group in the mITT Population

Table with similar format:

Table 18: Summary of Positive ADA Confirmation Assay Results by Time Point and Dose Cohort – Per-Protocol Population

Table 19: Anti-Drug Antibodies (ADA) Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Dose Cohort – mITT Population

| Time Point | Statistic | 3 mg/kg<br>EV68-228-N | 10 mg/kg<br>EV68-228-N | 30 mg/kg<br>EV68-228-N | Placebo |
|---|---|---|---|---|---|
| Day 1, | N | х | х | х | Х |
| Pre Dose | GMT | x.x | x.x | x.x | x.x |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Day 8 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 15 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 29 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 61 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 91 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 121 | N | | | | |
| C | GMT | | | | |
| | 95% CI | | | | |

Note: N=Number of participants in each group in the mITT Population.

Table 20: Anti-Drug Antibodies (ADA) Geometric Mean Titer (GMT) Results with 95% Confidence Intervals by Time Point and Dose Cohort – Per-Protocol Population

| Time Point | Statistic | 3 mg/kg<br>EV68-228-N<br>(N=X) | 10 mg/kg<br>EV68-228-N<br>(N=X) | 30 mg/kg<br>EV68-228-N<br>(N=X) | Placebo<br>(N=X) |
|---|---|---|---|---|---|
| Day 1, | N | х | х | x | х |
| Pre-Dose | GMT | x.x | x.x | X.X | X.X |
| | 95% CI | x.x, x.x | x.x, x.x | x.x, x.x | x.x, x.x |
| Day 8 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 15 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 29 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 61 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 91 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |
| Day 121 | N | | | | |
| | GMT | | | | |
| | 95% CI | | | | |

Note: N=Number of participants in each group in the Per-Protocol Population.

Table 21: Proportion of Participants with Detectable Anti-Drug Antibodies (ADA) with 95% Confidence Intervals by Time Point and Dose Cohort – mITT Population

[Implementation note: the Detectable Anti-Drug Antibodies means that in the confirmatory ADA assays, the results are positive.]

| Time Point | Statistics | 3 mg/kg<br>EV68-228-N | 10 mg/kg<br>EV68-228-N | 30 mg/kg<br>EV68-228-N | Placebo |
|---|---|---|---|---|---|
| Any time point | N | X | X | X | X |
| | n | х | х | x | X |
| | Proportion (95% CI) | x (x.xx, x.xx) | x (x.xx, x.xx) | x (x.xx, x.xx) | x (x.xx, x.xx) |
| Day 1, | N | х | х | x | X |
| Pre Dose | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 8 | N | x | Х | х | X |
| | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 15 | N | x | х | х | Х |
| | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 29 | N | x | х | х | X |
| | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 61 | N | х | Х | х | X |
| | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 121 | N | х | Х | х | X |
| | n | | | | |
| | Proportion (95% CI) | | | | |

Note: N=Number of participants in each group at the time point in the mITT Population.

Table 22: Proportion of Participants with Detectable Anti-Drug Antibodies (ADA) with 95% Confidence Intervals by Time Point and Dose Cohort – Per-Protocol Population

[Implementation note: the Detectable Anti-Drug Antibodies means that in the confirmatory ADA assays, the results are positive.]

| Time Point | Statistics | 3 mg/kg<br>EV68-228-N | 10 mg/kg<br>EV68-228-N | 30 mg/kg<br>EV68-228-N | Placebo |
|---|---|---|---|---|---|
| Any time point | N | х | X | X | Х |
| <b>-</b> | n | х | X | X | Х |
| | Proportion (95% CI) | x (x.xx, x.xx) | x (x.xx, x.xx) | x (x.xx, x.xx) | x (x.xx, x.xx) |
| Day 1, | N | х | X | X | Х |
| Pre Dose | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 8 | N | х | X | X | х |
| | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 15 | N | х | X | X | х |
| | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 29 | N | х | X | X | х |
| | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 61 | N | х | X | X | х |
| | n | | | | |
| | Proportion (95% CI) | | | | |
| Day 121 | N | х | X | X | х |
| | n | | | | |
| | Proportion (95% CI) | | | | |

Note: N=Number of participants in each group at the time point in the Per-Protocol Population.

#### **Safety Data** 14.3

## 14.3.1 Displays of Adverse Events

**Table 23: Overall Summary of Adverse Events** 

| | 3 mg/kg<br>EV68-228-N<br>(N=X) | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | Placebo<br>(N=X) | | All Participants who Received Active Product (N = x) | |
|---|---|---|---|---|---|---|---|---|---|---|
| Participants <sup>a</sup> with | n | % | n | % | n | % | n | % | n | % |
| At least one solicited adverse event | х | xx | х | xx | х | XX | х | XX | х | xx |
| At least one unsolicited adverse event | х | XX | х | xx | х | XX | х | XX | х | xx |
| At least one related unsolicited adverse event | х | XX | х | xx | х | XX | х | XX | х | xx |
| Mild (Grade 1) | х | XX | х | xx | х | XX | х | XX | х | xx |
| Moderate (Grade 2) | х | XX | х | xx | х | XX | х | XX | х | xx |
| Severe (Grade 3) | х | xxx | х | xx | х | XX | х | XX | х | xx |
| Life-threatening (Grade 4) | X | XX | х | xx | х | XX | х | XX | х | xx |
| Death (Grade 5) | | | | | | | | | | |
| At least one severe (Grade 3 or higher) unsolicited adverse event | | | | | | | | | | |
| Related | | | | | | | | | | |
| Unrelated | | | | | | | | | | |
| At least one serious adverse event <sup>b</sup> | | | | | | | | | | |
| At least one related, serious adverse event | | | | | | | | | | |
| At least one adverse event leading to early termination <sup>c</sup> | | | | | | | | | | |
| At least one unanticipated problem (UPs) | | | | | | | | | | |
| At least one medically attended adverse event (MAAEs) | | | | | | | | | | |
| At least one new onset chronic medical conditions (NOCMCs) | | | | | | | | | | |

Note: N=Number of participants in the Safety Population.

<sup>a</sup> Participants are counted once for each category regardless of the number of events.

<sup>&</sup>lt;sup>b</sup> A listing of Serious Adverse Events is included in Section 14.3.2.

<sup>&</sup>lt;sup>c</sup> As reported on the Adverse Event eCRF.

Table 24: Adverse Events Occurring in ≥ 5% of Participants in Any Dose Cohort by MedDRA System Organ Class and Preferred Term and Dose Cohort

[Implementation Note: This table will report both solicited and unsolicited AEs.]

| MedDRA System<br>Organ Class | MedDRA<br>Preferred | 1 | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | | Placebo<br>(N=X) | | | All Participants who Received<br>Active Product<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Term | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| Serious Adverse Even | ts | | | | | | | | | | | | | | • | |
| All | All | X | xx | X | X | xx | X | X | xx | x | X | XX | x | х | XX | х |
| SOC1 | All | | | | | | | | | | | | | | | |
| | PT1 | | | | | | | | | | | | | | | |
| | Etc. | | | | | | | | | | | | | | | |
| | All | | | | | | | | | | | | | | | |
| | PT1 | x | xx | x | x | xx | X | X | xx | х | x | xx | x | x | xx | х |
| Etc. | Etc. | | | | | | | | | | | | | | | |
| Other (Non-serious) A | dverse Events | | | | | | | | | | | | | | | |
| All | All | x | xx | X | X | xx | x | X | xx | x | x | xx | x | х | xx | x |
| SOC1 | All | x | xx | x | x | xx | x | X | xx | х | x | xx | x | x | xx | х |
| | PT1 | | | | | | | | | | | | | | | |
| | Etc. | | | | | | | | | | | | | | | |
| Etc | Etc | | | | | | | | | | | | | | | |

Notes: N=Number of participants in the Safety Population. n=Number of participants reporting an event. Events=Total frequency of events reported.

### **14.3.1.1** Solicited Adverse Events

Table 25: Number and Percentage of Participants Experiencing Solicited Events with 95% Confidence Intervals by Symptom and Dose Cohort

| | 3 mg/kg<br>EV68-228-N<br>(N=X) | | 10 mg/kg<br>EV68-228-N<br>(N=X) | | | 30 mg/kg<br>EV68-228-N<br>(N=X) | | | | Placebo<br>(N=X) | ) | All Participants who<br>Received Active<br>Product<br>(N=X) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI | n | % | 95%<br>CI |
| Any Symptom | х | xx | X.X,<br>X.X | х | xx | x.x,<br>x.x | x | xx | x.x,<br>x.x | x | xx | x.x,<br>x.x | X | xx | X.X,<br>X.X |
| Headache | | | | | | | | | | | | | | | |
| Rash | | | | | | | | | | | | | | | |
| Nausea | | | | | | | | | | | | | | | |
| Vomiting | | | | | | | | | | | | | | | |
| Diarrhea | | | | | | | | | | | | | | | |
| Fatigue (Tiredness) | | | | | | | | | | | | | | | |
| Myalgia (Body<br>aches/Muscular pain) | | | | | | | | | | | | | | | |

Notes: N=Number of participants in the Safety Population. 95% CI=Clopper-Pearson confident interval.
Table 26: Comparison of the Proportion of Participants Experiencing Solicited Events by Dose Cohort

| Symptom | Statistic | 3 mg/kg<br>EV68-228-N<br>(N=X) | 10 mg/kg<br>EV68-228-N<br>(N=X) | 30 mg/kg<br>EV68-228-N<br>(N=X) | Placebo<br>(N=X) |
|---|---|---|---|---|---|
| Any Symptom | Proportion | x.xx | x.xx | x.xx | x.xx |
| | 95% CI (for proportion) <sup>a</sup> | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | x.xx | X.XX | X.XX | - |
| | 95% CI (for difference) <sup>b</sup> | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | - |
| Headache | Proportion | x.xx | x.xx | x.xx | x.xx |
| | 95% CI (for proportion) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | x.xx | x.xx | x.xx | - |
| | 95% CI (for difference) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | - |
| Rash | Proportion | x.xx | x.xx | x.xx | x.xx |
| | 95% CI (for proportion) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | x.xx | x.xx | x.xx | - |
| | 95% CI (for difference) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | - |
| Nausea | Proportion | x.xx | x.xx | x.xx | x.xx |
| | 95% CI (for proportion) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | x.xx | x.xx | x.xx | - |
| | 95% CI (for difference) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | - |
| Vomiting | Proportion | x.xx | x.xx | x.xx | x.xx |
| | 95% CI (for proportion) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | x.xx | x.xx | x.xx | - |
| | 95% CI (for difference) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | - |
| Diarrhea | Proportion | x.xx | x.xx | x.xx | x.xx |
| | 95% CI (for proportion) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | x.xx | x.xx | x.xx | - |
| | 95% CI (for difference) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | - |
| Fatigue | Proportion | x.xx | x.xx | x.xx | x.xx |
| (Tiredness) | 95% CI (for proportion) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | x.xx | x.xx | x.xx | - |
| | 95% CI (for difference) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | - |
| Myalgia | Proportion | x.xx | X.XX | x.xx | x.xx |
| (Body aches/Muscular pain) | 95% CI (for proportion) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx |
| | Difference | x.xx | X.XX | X.XX | - |
| | 95% CI (for difference) | x.xx, x.xx | x.xx, x.xx | x.xx, x.xx | - |

Note: N=Number of participants in the Safety Population.

<sup>&</sup>lt;sup>a</sup>95% CI=Clopper-Pearson confidence interval.

b95% CI=Wald confidence interval.

Table 27: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Maximum Severity, and Dose Cohort

| | | EV68- | g/kg<br>-228-N<br>=X) | EV68- | ng/kg<br>-228-N<br>=X) | EV68- | ng/kg<br>-228-N<br>=X) | | cebo<br>=X) | who R<br>Active | ticipants<br>eceived<br>Product<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % |
| Any Symptom | None | X | XX | X | xx | x | xx | x | xx | Х | XX |
| | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| | Life-threatening | | | | | | | | | | |
| Headache | None | X | xx | х | xx | х | xx | х | xx | х | XX |
| | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| | Life-threatening | | | | | | | | | | |
| Rash | None | X | xx | х | xx | х | xx | х | xx | х | XX |
| | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| | Life-threatening | | | | | | | | | | |
| Nausea | None | X | xx | х | xx | х | xx | х | xx | х | XX |
| | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| | Life-threatening | | | | | | | | | | |
| Vomiting | None | X | xx | х | xx | х | xx | х | xx | х | XX |
| | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| | Life-threatening | | | | | | | | | | |
| Diarrhea | None | X | xx | X | XX | X | xx | X | XX | X | XX |
| | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| | Life-threatening | | | | | | | | | | |
| Fatigue | None | X | xx | X | XX | X | xx | X | XX | X | XX |
| (Tiredness) | Mild | | | | | | 1 | | 1 | | |

Table 27: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Maximum Severity, Dose, and Dose Cohort (continued)

| | | EV68- | g/kg<br>-228-N<br>=X) | EV68- | ng/kg<br>-228-N<br>=X) | EV68- | ng/kg<br>-228-N<br>=X) | | cebo<br>=X) | who R<br>Active | ticipants<br>eceived<br>Product<br>=X) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Symptom | Severity | n | % | n | % | n | % | n | % | n | % |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| | Life-threatening | | | | | | | | | | |
| Myalgia (Body | None | X | xx | x | xx | X | xx | x | xx | x | xx |
| aches/Muscular pain) | Mild | | | | | | | | | | |
| | Moderate | | | | | | | | | | |
| | Severe | | | | | | | | | | |
| | Life-threatening | | | | | | | | | | |

Notes: N=Number of participants in the Safety Population. Severity is the maximum severity reported over all solicited symptoms post dosing for each participant.

Table 28: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – 3 mg/kg EV68-228-N

| | | | | | 3 mg/kg E<br>(N: | V68-228-I<br>=X) | N | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Da | ıy 1 | Da | ny 2 | Da | ay 3 | Ongoin<br>Da | g After<br>y 3 |
| Symptom | Severity | n | % | n | % | n | % | n | % |
| Any Symptom | None | X | XX | X | XX | X | XX | X | XX |
| | Mild | | | | | | | | |
| | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Life-threatening | | | | | | | | |
| | Not Reported | | | | | | | | |
| Headache | None | | | | | | | | |
| | Mild | | | | | | | | |
| | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Life-threatening | | | | | | | | |
| | Not Reported | | | | | | | | |
| Rash | None | | | | | | | | |
| | Mild | | | | | | | | |
| | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Life-threatening | | | | | | | | |
| | Not Reported | | | | | | | | |
| Nausea | None | | | | | | | | |
| | Mild | | | | | | | | |
| | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Life-threatening | | | | | | | | |
| | Not Reported | | | | | | | | |
| Vomiting | None | | | | | | | | |
| | Mild | | | | | | | | |
| | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Life-threatening | | | | | | | | |
| | Not Reported | | | | | | | | |
| Diarrhea | None | | | | | | | | |
| | Mild | | | | | | | | |
| | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Life-threatening | | | | | | | | |
| | Not Reported | | | | | 1 | | | |
| Fatigue | None | | | | | | | | |
| 5 | Mild | | | | | | | | |
| | Moderate | | | | | 1 | | | |
| | Moderate | | | 1 | | | | | |

Table 28:Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing – 3 mg/kg EV68-228-N (continued)

| | | | | | 3 mg/kg E<br>(N= | V68-228-N<br>=X) | I | | |
|---|---|---|---|---|---|---|---|---|---|
| | | Da | ny 1 | Da | ny 2 | Da | y 3 | Ongoir<br>Da | g After<br>y 3 |
| Symptom | Severity | n | % | n | % | n | % | n | % |
| | Severe | | | | | | | | |
| | Life-threatening | | | | | | | | |
| | Not Reported | | | | | | | | |
| Myalgia | None | | | | | | | | |
| | Mild | | | | | | | | |
| | Moderate | | | | | | | | |
| | Severe | | | | | | | | |
| | Life-threatening | | | | | | | | |
| | Not Reported | | | | | | | | |

Notes: N=Number of participants in the Safety Population. Severity is the maximum severity reported post dosing for each participant for each day.

#### Tables with similar format:

- Table 29: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing 10 mg/kg EV68-228-N
- Table 30: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing 30 mg/kg EV68-228-N
- Table 31: Number and Percentage of Participants Experiencing Solicited Events by Symptom, Severity, and Day Post Dosing Placebo

#### 14.3.1.2 **Unsolicited Adverse Events**

Summary of Unsolicited Adverse Events by MedDRA System Organ Class, High Level Group Term and Preferred Term and Table 32: **Dose Cohort** 

| MedDRA | MedDRA<br>High Level<br>Group | MedDRA | 3 r | | V68-228<br>=X) | 8-N | 10 | mg/kg I<br>(N: | EV68-22<br>=X) | 28-N | 30 1 | mg/kg I<br>(N: | EV68-22<br>=X) | 28-N | | | cebo<br>=X) | | | ived Ac | ipants w<br>tive Pro<br>=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System<br>Organ Class | Term | Preferred<br>Term | n | % | 95%<br>CI <sup>a</sup> | Even<br>ts | n | % | 95%<br>CI <sup>a</sup> | Event<br>s | n | % | 95%<br>CI <sup>a</sup> | Event<br>s | n | % | 95%<br>CI <sup>a</sup> | Event<br>s | n | % | 95%<br>CI <sup>a</sup> | Even<br>ts |
| Any SOC | Any HLGT | Any PT | X | xx | xx,<br>xx | x | X | xx | xx,<br>xx | x | X | xx | xx,<br>xx | x | x | xx | xx,<br>xx | х | x | xx | xx,<br>xx | x |
| [SOC 1] | Any HLGT | Any PT | | | | | | | | | | | | | | | | | | | | |
| | HLGT1 | Any PT | | | | | | | | | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| | HLGT2 | Any PT | | | | | | | | | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| [SOC 2] | Any HLGT | Any PT | | | | | | | | | | | | | | | | | | | | |
| | HLGT1 | Any PT | | | | | | | | | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | | | | | | | | | |
| | HLGT2 | Any PT | | | | | | | | | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | | | | | | | | | |

Notes: N=Number of participants in the Safety Population. This table presents the number and percentage of participants. A participant is only counted once per PT. 

<sup>a</sup> The 95% CI of the proportion will be calculated using Clopper-Pearson (Exact) methodology from a binomial distribution.

Table 33: Unsolicited Adverse Events by MedDRA System Organ Class, High Level Group Term and Preferred Term, Maximum Severity, and Dose Cohort

| MedDRA System | MedDRA<br>High Level<br>Group | MedDRA | | EV68 | ng/kg<br>3-228-N<br>(=X) | | ng/kg<br>-228-N<br>=X) | EV68 | mg/kg<br>3-228-N<br>(=X) | _ | icebo<br>(=X) | Active | s who Received<br>Product<br>= X) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Organ Class | Term | Preferred Term | Severity | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any HLGT | Any PT | Any Severity | X | xx | X | XX | X | xx | X | xx | X | xx |
| | | | Mild | X | XX | X | XX | X | XX | X | xx | x | xx |
| | | | Moderate | X | XX | X | XX | X | XX | X | xx | X | xx |
| | | | Severe | X | XX | X | XX | х | xx | X | XX | X | xx |
| | | | Life-threatening | X | xx | X | XX | х | xx | X | xx | x | xx |
| SOC 1 | Any HLGT | Any PT | Any Severity | Х | XX | Х | XX | х | xx | х | XX | х | xx |
| | | | Mild | х | xx | х | XX | х | xx | х | xx | х | xx |
| | | | Moderate | х | xx | Х | XX | х | xx | х | xx | х | xx |
| | | | Severe | х | xx | Х | XX | х | xx | х | xx | х | xx |
| | | | Life-threatening | х | XX | Х | XX | х | xx | х | XX | х | xx |
| | HLGT1 | PT1 | Any Severity | х | xx | Х | XX | х | xx | х | xx | х | xx |
| | | | Mild | х | xx | Х | XX | х | xx | х | xx | х | xx |
| | | | Moderate | х | XX | х | XX | х | xx | х | XX | х | xx |
| | | | Severe | х | XX | х | XX | х | xx | х | XX | х | xx |
| | | | Life-threatening | х | XX | х | XX | х | xx | х | XX | х | xx |
| | | PT2 | Any Severity | х | XX | х | XX | х | XX | х | XX | х | xx |
| | | | Mild | х | XX | х | XX | х | XX | х | XX | х | xx |
| | | | Moderate | х | XX | х | XX | х | XX | х | XX | х | xx |
| | | | Severe | х | XX | х | XX | х | XX | х | XX | х | xx |
| | | | Life-threatening | Х | xx | Х | XX | х | xx | Х | xx | х | xx |

Notes: N=Number of participants in the Safety Population. This table presents the number and percentage of participants. A participant is only counted once by the maximal severity per PT.

Table 34: Unsolicited Adverse Events by MedDRA System Organ Class, High Level Group Term and Preferred Term, Maximum Severity, Relationship, and Dose Cohort

| | | | | | EV68 | g/kg<br>-228-N<br>=X) | 1 | | EV68 | ng/kg<br>-228-N<br>=X) | V | | EV68 | ng/kg<br>-228-N<br>=X) | J. | | | cebo<br>=X) | | v | II Part<br>who Roctive I | eceive | ed |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| MedDRA<br>System | MedDRA High<br>Level Group | MedDRA<br>Preferred | | Rel | ated | | ot<br>ated | Rel | ated | | ot<br>ated | Rel | ated | | ot<br>ated | Rel | ated | | ot<br>ated | Rel | ated | | lot<br>ated |
| Organ Class | Term | Term | Severity | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % | n | % |
| Any SOC | Any HLGT | Any PT | Any Severity | Х | XX | X | XX | Х | XX | Х | XX | Х | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | | | Mild | X | xx | X | XX | Х | XX | Х | XX | Х | XX | X | XX | X | XX | X | XX | X | xx | X | XX |
| | | | Moderate | Х | XX | X | XX | Х | XX | Х | XX | Х | XX | X | XX | X | XX | X | XX | X | XX | X | XX |
| | | | Severe | X | xx | X | XX | Х | XX | Х | XX | Х | XX | X | XX | X | XX | X | XX | X | xx | X | XX |
| | | | Life-threatening | X | xx | X | XX | Х | XX | Х | XX | Х | XX | X | XX | X | XX | X | XX | X | xx | X | XX |
| SOC 1 | Any HLGT | Any PT | Any Severity | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx |
| | | | Mild | X | xx | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx | X | XX |
| | | | Moderate | X | xx | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx | X | XX |
| | | | Severe | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx | X | xx |
| | | | Life-threatening | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx | X | xx |
| | HLGT1 | Any PT | Any Severity | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx | X | xx |
| | | | Mild | X | xx | x | XX | X | XX | X | XX | X | XX | Х | XX | X | xx | x | XX | X | xx | x | XX |
| | | | Moderate | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx | X | xx |
| | | | Severe | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx | X | xx |
| | | | Life-threatening | X | xx | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx | X | xx |
| | | PT 1 | Any Severity | X | xx | x | XX | X | XX | X | XX | X | XX | X | XX | X | XX | x | XX | X | xx | X | XX |
| | | | Mild | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | Х | XX | X | XX | Х | xx |
| | | | Moderate | X | XX | x | XX | X | XX | X | XX | X | XX | X | XX | х | xx | X | XX | X | XX | х | xx |
| | | | Severe | X | XX | x | XX | X | XX | X | XX | X | XX | X | XX | х | xx | X | XX | X | XX | х | xx |
| | | | Life-threatening | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | xx |

Table 34: Unsolicited Adverse Events by MedDRA System Organ Class, High Level Group Term and Preferred Term, Maximum Severity, Relationship, and Dose Cohort (continued)

| PT 2 | Any Severity | X | XX | X | XX | X | XX | x | XX | X | XX | X | XX | X | XX | x | xx | X | XX | X | xx |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Mild | X | XX | X | XX | X | xx | X | XX | х | XX | X | XX | X | XX | х | XX | X | XX | X | xx |
| | Moderate | X | XX | X | XX | X | xx | X | XX | х | XX | X | XX | X | XX | х | XX | X | XX | X | xx |
| | Severe | X | XX | X | XX | X | xx | X | XX | х | XX | X | XX | X | XX | х | XX | X | XX | X | xx |
| | Life-threatening | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX | X | XX |

Notes: N=Number of participants in the Safety Population. This table presents the number and percentage of participants. A participant is only counted once by the maximum severity per PT.

Table 35: Related Unsolicited Adverse Events Post Dosing by MedDRA System Organ Class, High Level Group Term and Preferred Term, and Dose Cohort

| MedDRA<br>System<br>Organ | MedDRA<br>High Level<br>Group Term | MedDRA | 3 mg | /kg EV68-<br>(N=X) | -228-N | 10 m | g/kg EV68<br>(N=X) | | 30 mg | /kg EV68<br>(N=X) | -228-N | | Placebo<br>(N=X) | | | articipanted Active (N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Class | | Preferred Term | n | % | Events | n | % | Events | n | % | Events | n | % | Events | n | % | Events |
| Any SOC | Any HLGT | Any PT | X | XX | X | X | XX | x | X | XX | X | X | XX | X | X | XX | x |
| [SOC 1] | Any HLGT | Any PT | | | | | | | | | | | | | | | |
| | HLGT1 | Any PT | | | | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | | | | |
| | HLGT2 | Any PT | | | | | | | | | | | | | | | |
| | | [PT 1] | | | | | | | | | | | | | | | |
| | | [PT 2] | | | | | | | | | | | | | | | |

Notes: N=Number of participants in the Safety Population. This table presents the number and percentage of participants. A participant is only counted once per PT.

## 14.3.2 Listing of Deaths, Other Serious and Significant Adverse Events

 Table 36:
 Listing of Serious Adverse Events

| Adverse<br>Event | No. of<br>Days Post<br>Dose<br>(Duration) | No. of<br>Days Post<br>Dose the<br>Event<br>Became<br>Serious | Reason<br>Reported<br>as an SAE | Severity | Relationsh<br>ip to<br>Study<br>Treatment | If Not<br>Related,<br>Alternativ<br>e Etiology | Action<br>Taken<br>with Study<br>Treatment | Participant<br>Discontinu<br>ed Due to<br>AE | MAAE/<br>NOCMC/<br>UP? | Outcome | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>High<br>Level<br>Group<br>Term | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose Cohort | t:, Participant | ID:, AE Num | ber: | | | | | | | | | | |
| <b>Comments:</b> | | | | | | | | | | | | | |
| Dose Cohort | t:, Participant | ID:, AE Num | ber: | | | | | | | | | | |
| Comments: | | | | | | | | | | | | | |

## Table 37: Listing of Non-Serious, Unsolicited, Moderate or Severe Adverse Events

[Implementation note: All Non-Serious AEs, which are greater than grade 2, will be included.]

| Adverse<br>Event | No. of Days<br>Post Dose<br>(Duration) | Severity | Relationship<br>to Study<br>Treatment | If Not<br>Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Participant<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ<br>Class | MedDRA<br>High Level<br>Group Term | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|
| Dose Cohort:, P | articipant ID:, A | E Number: | | | | | | | | |
| Comments: | | | | | • | | • | | | |
| Dose Cohort:, P | articipant ID:, A | E Number: | | | | | | | | |
| Comments: | | | | | | | | | | |

## **Table 38:** Listing of Other Significant Adverse Events

[Implementation Note: Other Significant Adverse Events include New Onset Chronic Medical Conditions (NOCMC), Medically Attended Adverse Events (MAAEs).]

| Adverse<br>Event<br>Dose Cohort | No. of Days<br>Post Dose<br>(Duration)<br>:, Participant ID: | Severity<br>AE Number: | Relationship<br>to Study<br>Treatment | If Not Related,<br>Alternative<br>Etiology | Action Taken<br>with Study<br>Treatment | Participant<br>Discontinued<br>Due to AE | Outcome | MAAE/<br>NOCMC/<br>UP? | MedDRA<br>System<br>Organ<br>Class | MedDRA<br>High<br>Level<br>Group<br>Term | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Comments: | | | | | | | | | | | |

#### **Table 39:** Listing of Participant-Specific Unanticipated Problems (UPs)

[Implementation note: "Study Day" is relative to treatment administration; the day of treatment administration is Day 1, and the day prior to treatment administration is Day -1.

If event is an AE, display "Yes" followed by the AE description and number separated by a semicolon in parentheses.

If event is a PD, display "Yes" followed by the deviation description and number separated by a semicolon in parentheses.

If there are no comments, display "None" in the "Comments" column. If there are no comments for any UPs in the listing, remove the "Comments" column. If the comments are too long to display in the "Comments" column, the format of this table may be updated to remove the "Comments" column.

Sort by Dose Cohort, Participant ID, and UP Number.]

| Dose Cohort | Participant<br>ID | UP number | Event<br>Description | Event<br>Outcome | Study Day of<br>Site<br>Awareness | Study Day<br>Reported to<br>Sponsor/DCC | Study Day<br>Reported<br>to IRB | Is the event an AE (AE Description; Number) | Is the event an PD (DV Description; Number) | Comments |
|---|---|---|---|---|---|---|---|---|---|---|
| 3 mg/kg<br>EV68-228-N | ZZZ.XXXXX | xxx | [description] | [outcome] | х | Х | х | No | No | |
| 10 mg/kg<br>EV68-228-N | | | | | | | | Yes<br>([description];<br>XXX) | Yes<br>([description];<br>XXX) | |
| 30 mg/kg<br>EV68-228-N | | | | | | | | | | |

Abbreviations: UP = Unanticipated Problem; DCC - Data Coordinating Center; IRB = Institutional Review Board; AE = Adverse Event; PD = Protocol Deviation; DV = Deviation.

## **Table 40:** Listing of Non-Participant Specific Unanticipated Problems (UPs)

[implementation note:

If event is a PD, display "Yes" followed by the deviation description and number separated by a semicolon in parentheses.

If there are no comments, display "None" in the "Comments" column. If there are no comments for any UPs in the listing, remove the "Comments" column. If the comments are too long to display in the "Comments" column, the format of this table may be updated to remove the "Comments" column.

Sort by Site and UP Number]

| Site | UP<br>number | Event<br>Description | Event<br>Outcome | Event Date | Date of Site<br>Awareness | Study Day<br>Reported to<br>Sponsor/DCC | Study Day<br>Reported to IRB | Is the event an PD (DV Description Number) | Comments |
|---|---|---|---|---|---|---|---|---|---|
| University of Maryland | xxx | [description] | [outcome] | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | DDMMMYYYY | No | |
| Vanderbilt<br>University | | | | | | | | Yes ([description]; XXX) | |

Abbreviations: UP = Unanticipated Problem; DCC - Data Coordinating Center; IRB = Institutional Review Board; AE = Adverse Event; PD = Protocol Deviation; DV = Deviation.

## 14.3.3 Narratives of Deaths, Other Serious and Significant Adverse Events

Not included in SAP, but this is a placeholder for the CSR.

## 14.3.4 Abnormal Laboratory Value Listings (by Participant)

## Table 41: Listing of Abnormal Laboratory Results – Chemistry

| Dose Cohort | Participant<br>ID | Sex | Age (years) | Planned Time<br>Point | Actual Study<br>Day | Laboratory<br>Parameter<br>(Units) | Result<br>(Severity) | Relationship<br>to Treatment | If Not<br>Related,<br>Alternate<br>Etiology | Clinically<br>Significant? | Participation Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

 Table 42:
 Listing of Abnormal Laboratory Results – Hematology

| Dose<br>Cohort | Participant<br>ID | Sex | Age<br>(years) | Planned<br>Time Point | Actual<br>Study Day | Laboratory Parameter (Units) | Result<br>(Severity) | Relationship to<br>Treatment | If Not Related,<br>Alternate<br>Etiology | Clinically<br>Significant? | Participant Discontinued Due to Result? |
|---|---|---|---|---|---|---|---|---|---|---|---|

 Table 43:
 Listing of Abnormal Laboratory Results – Hypersensitivity

| Dose Cohort | Participant<br>ID | Sex | Age<br>(years) | Planned Time Point | Actual Study<br>Day | Parameter | Units | Result | Clinically<br>Significant? |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Baseline/ Onset of symptom/ 2 or more hours after onset/ Resolution of symptom | | Complement Component 3/ Complement Component 4/ CH50/ Immunoglobin E/ Serum Tryptase | | x | CS/NCS |

## 14.3.5 Displays of Laboratory Results

## 14.3.5.1 Chemistry Results

## Table 44: Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Chemistry Parameter

| Any Chemistry | | | No | one | Mil<br>Grad | | | derate/<br>rade 2 | Seve<br>Grae | | Life-thre<br>Grae | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | 3 mg/kg EV68-228-N | х | Х | xx | х | xx | х | XX | х | xx | х | xx |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 2 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 3 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 8 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 29 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Table 44: Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort - Any Chemistry Parameter (continued)

| Any Chemistry | | | No | one | Mil<br>Grad | | | derate/<br>cade 2 | Seve<br>Grad | | Life-three<br>Grad | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| j | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Notes: The "Max Severity Post Baseline" rows indicate the maximum severity experienced by each participant at any time point post baseline, including unscheduled assessments. N=Number of participants in the Safety Population.

Table 45: Laboratory Results by Parameter Time Point, and Dose Cohort – Chemistry: Creatinine

| | | | N | one | Mi<br>Gra | ild/<br>de 1 | | derate/<br>rade 2 | | vere/<br>ade 3 | Life-thre<br>Grad | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Creatinine Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | 3 mg/kg EV68-228-N | х | X | xx | X | xx | х | XX | х | XX | х | xx |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 2 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 3 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 8 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 29 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Table 45: Laboratory Results by Parameter Time Point, and Dose Cohort – Chemistry: Creatinine (continued)

| | | | No | one | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | vere/<br>ade 3 | Life-three<br>Grad | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| <b>Creatinine Time Point</b> | Dose Cohort | N | n | n % | % | n | % | n | % | n | % |
| Max Severity Post Baseline | 3 mg/kg EV68-228-N | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | |
| | Placebo | | | | | | | | | | |

Notes: The "Max Post Baseline" rows indicate the maximum severity experienced by each participant at any time point post baseline, including unscheduled assessments. N=Number of participants in the Safety Population.

#### Tables with similar format:

Table 46: Laboratory Results by Parameter Time Point, and Dose Cohort – Total Bilirubin

Table 47: Laboratory Results by Parameter Time Point, and Dose Cohort – ALT

Table 48: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Chemistry Parameter

| Any Chemistry | | | No | one | | ild/<br>nde 1 | | lerate/<br>ade 2 | | vere/<br>ade 3 | | eatening/<br>ade 4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | 3 mg/kg EV68-228-N | х | Х | xx | Х | xx | X | xx | X | xx | х | xx |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 2 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 3 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 8 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 29 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Table 48: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Chemistry Parameter (continued)

| Any Chemistry | | | No | one | | ild/<br>de 1 | Mode<br>Gra | erate/<br>de 2 | | rere/<br>ade 3 | | eatening/<br>ide 4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| · · · · · | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Notes: The "Max Post Baseline" rows indicate the maximum severity experienced by each participant at any time point post baseline, including unscheduled assessments. N=Number of participants in the Safety Population

### Tables with similar format:

Table 49: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Creatinine

Table 50: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Total

Bilirubin

Table 51: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – ALT

Table 52: Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – Creatinine

| <b>Time Point</b> | Dose Cohort | N | Mean | <b>Standard Deviation</b> | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | 3 mg/kg EV68-228-N | х | XX.X | XX.X | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 2 | 3 mg/kg EV68-228-N | х | XX.X | XX.X | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 2, Change from Baseline | 3 mg/kg EV68-228-N | х | XX.X | XX.X | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 3 | 3 mg/kg EV68-228-N | х | XX.X | XX.X | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 3, Change from Baseline | 3 mg/kg EV68-228-N | х | XX.X | XX.X | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 8 | 3 mg/kg EV68-228-N | Х | XX.X | xx.x | XX.X | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 8, Change from Baseline | 3 mg/kg EV68-228-N | Х | XX.X | xx.x | XX.X | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 29 | 3 mg/kg EV68-228-N | х | XX.X | xx.x | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 29, Change from Baseline | 3 mg/kg EV68-228-N | х | XX.X | xx.x | XX.X | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |

Note: N=Number of participants in the Safety Population with non-missing values at respective visit.

## Tables with similar format:

Table 53: Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – Total

Bilirubin

Table 54: Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – ALT

## 14.3.5.2 Hematology Results

## Table 55: Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Hematology Parameter

| Any Hematology | | | No | one | | ild/<br>ade 1 | | erate/<br>ide 2 | Seve<br>Grae | | | reatening/<br>rade 4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | 3 mg/kg EV68-228-N | х | Х | xx | Х | xx | х | xx | х | XX | х | XX |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 2 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 3 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 8 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 29 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Table 55: Laboratory Results by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Hematology Parameter (continued)

| Any Hematology | | | No | one | | ld/<br>de 1 | | erate/<br>de 2 | Seve<br>Grad | | | reatening/<br>ade 4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Parameter Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Notes: The "Max Post Baseline" rows indicate the maximum severity experienced by each participant at any time point post baseline, including unscheduled assessments. N=Number of participants in the Safety Population.

#### Tables with similar format:

| Table 56: | Laboratory | Results by | Parameter. | Maximum | Severity, | Time Point, | and Dose Coho | rt – Hemoglobin |
|---|---|---|---|---|---|---|---|---|

# Table 60: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Hematology Parameter

| | | | N | one | | ild/<br>ade 1 | | lerate/<br>ade 2 | Severe/<br>Grade 3 | | Life-threatening/<br>Grade 4 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | 3 mg/kg EV68-228-N | х | х | xx | X | xx | x | xx | Х | xx | х | XX |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 2 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 3 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 8 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 29 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Table 60: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Any Hematology Parameter

| | | | None | | Mild/<br>Grade 1 | | Moderate/<br>Grade 2 | | Severe/<br>Grade 3 | | Life-threatening/<br>Grade 4 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Max Severity Post Baseline | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Notes: The "Max Post Baseline" rows indicate the maximum severity experienced by each participant at any time point post baseline, including unscheduled assessments. N=Number of participants in the Safety Population.

#### Tables with similar format:

Table 61: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Hemoglobin

Table 62: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – WBC – Low

Table 63: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – WBC – High

Table 64: Laboratory Results Related to Study Treatment by Parameter, Maximum Severity, Time Point, and Dose Cohort – Platelets

Table 65: Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – Hemoglobin

| Time Point | Dose Cohort | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Baseline | 3 mg/kg EV68-228-N | x | xx.x | XX.X | XX.X | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 2 | 3 mg/kg EV68-228-N | x | XX.X | XX.X | XX.X | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 2, Change from Baseline | 3 mg/kg EV68-228-N | x | xx.x | XX.X | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 3 | 3 mg/kg EV68-228-N | х | XX.X | XX.X | XX.X | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 3, Change from Baseline | 3 mg/kg EV68-228-N | x | XX.X | XX.X | XX.X | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 8 | 3 mg/kg EV68-228-N | x | xx.x | XX.X | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 8, Change from Baseline | 3 mg/kg EV68-228-N | x | xx.x | XX.X | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |
| Day 29 | 3 mg/kg EV68-228-N | х | XX.X | XX.X | XX.X | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |

Table 65: Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – Hemoglobin (continued)

| Time Point | Dose Cohort | N | Mean | Standard<br>Deviation | Median | Min, Max |
|---|---|---|---|---|---|---|
| Day 29, Change from Baseline | 3 mg/kg EV68-228-N | X | XX.X | xx.x | xx.x | xx.x, xx.x |
| | 10 mg/kg EV68-228-N | | | | | |
| | 30 mg/kg EV68-228-N | | | | | |
| | Placebo | | | | | |

Note: N=Number of participants in the Safety Population with non-missing values at respective visit.

#### Tables with similar format:

Table 66: Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – WBC

Table 67: Laboratory Summary Statistics by Parameter, Time Point, and Dose Cohort – Platelets

## 14.3.6 Displays of Vital Signs

## Table 68: Vital Signs by Maximum Severity, Time Point, and Dose Cohort – Any Assessment

| | | | N | one | | ild/<br>ade 1 | | lerate/<br>ade 2 | | vere/<br>ade 3 | | eatening/<br>ide 4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | Dose Cohort | N | n | % | n | % | n | % | n | % | n | % |
| Baseline | 3 mg/kg EV68-228-N | х | x | xx | X | xx | x | xx | х | XX | X | xx |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| 15 Min After start of | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| Infusion | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| End of Infusion | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| 1 Hour After End of | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| Infusion | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 2 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |
| Day 3 | 3 mg/kg EV68-228-N | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | |

Table 68: Vital Signs by Maximum Severity, Time Point, and Dose Cohort – Any Assessment (continued)

| | Dose Cohort | David David | | N | one | | ild/<br>ade 1 | | erate/<br>ide 2 | Sev<br>Gra | ere/<br>de 3 | | eatening/<br>de 4 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time Point | | N | n | % | n | % | n | % | n | % | n | % | |
| Day 8 | 3 mg/kg EV68-228-N | | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | | |
| Day 15 | 3 mg/kg EV68-228-N | | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | | |
| Day 29 | 3 mg/kg EV68-228-N | | | | | | | | | | | | |
| | 10 mg/kg EV68-228-N | | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | | |
| Max Severity Post | 3 mg/kg EV68-228-N | | | | | | | | | | | | |
| Baseline | 10 mg/kg EV68-228-N | | | | | | | | | | | | |
| | 30 mg/kg EV68-228-N | | | | | | | | | | | | |
| | Placebo | | | | | | | | | | | | |

Notes: The "Max Severity Post Baseline" rows indicate the maximum severity experienced by each participant at any time point post baseline, including unscheduled assessments. N = Number of participants in the Safety Population.

#### Tables with similar format:

- Table 69: Vital Signs by Assessment, Maximum Severity, Time Point, and Dose Cohort Body Temperature
- Table 70: Vital Signs by Assessment, Maximum Severity, Time Point, and Dose Cohort Pulse: High
- Table 71: Vital Signs by Assessment, Maximum Severity, Time Point, and Dose Cohort Pulse: Low
- Table 72: Vital Signs by Assessment, Maximum Severity, Time Point, and Dose Cohort Systolic Blood Pressure: High
- Table 73: Vital Signs by Assessment, Maximum Severity, Time Point, and Dose Cohort Systolic Blood Pressure: Low
- Table 74: Vital Signs by Assessment, Maximum Severity, Time Point, and Dose Cohort Diastolic Blood Pressure: High

Table 75: Summary of Post Dose ECG Change in Overall Interpretations from Baseline by Dose Cohort and Time Point

| Time Point | Change from Baseline in ECG Interpretation | 3 mg/kg<br>EV68-228-N | 10 mg/kg<br>EV68-228-N | 30 mg/kg<br>EV68-228-N | Placebo | All Participants |
|---|---|---|---|---|---|---|
| 1 Hour post | N | x | X | x | x | x |
| Infusion | Normal at Both Times, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Normal to Abnormal, NCS, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Normal to Abnormal, CS, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Abnormal, NCS at Both Times, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Abnormal, NCS to Abnormal, CS, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Abnormal, NCS to Normal, n (%) | x(x) | x(x) | x(x) | x(x) | x(x) |
| Day 2 | N | x | X | x | х | x |
| | Normal at Both Times, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Normal to Abnormal, NCS, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Normal to Abnormal, CS, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Abnormal, NCS at Both Times, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Abnormal, NCS to Abnormal, CS, n (%) | x (x) | x (x) | x (x) | x (x) | x (x) |
| | Abnormal, NCA to Normal, n (%) | x(x) | x(x) | x(x) | x(x) | x(x) |

Notes: N=Number of participants in the Safety Population with ECG measurements at the time points indicated. NCS=Not clinically significant. CS=Clinically significant.
## 14.4 Summary of Concomitant Medications

Table 76: Number and Percentage of Participants with Prior and Concurrent Medications by WHO Drug Classification and Dose Cohort

| WHO Drug Code<br>Level 1, | WHO Drug Code<br>Level 2, | Level 2, | | EV68- | ng/kg<br>-228-N<br>=X) | EV68- | ng/kg<br>-228-N<br>=X) | Placebo<br>(N=X) | | All Participants<br>(N=X) | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Anatomic Group | Therapeutic Subgroup | n | % | n | % | n | % | n | % | n | % |
| Any Level 1 Codes | Any Level 2 Codes | X | xx | X | XX | X | XX | X | xx | x | xx |
| [ATC Level 1 - 1] | Any [ATC 1 – 1] | | | | | | | | | | |
| | [ATC 2 - 1] | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | |
| [ATC Level 1 – 2] | [ATC 2 - 1] | | | | | | | | | | |
| | [ATC 2 - 2] | | | | | | | | | | |
| | [ATC 2 - 3] | | | | | | | | | | |

Notes: N=Number of participants enrolled in each group. n=Number of participants reporting taking at least one medication in the specific WHO Drug Class.

#### 14.5 EV68-228-N Serum Concentrations and PK Parameters

Table 77: Individual Statistics of Serum EV68-228-N Concentrations by Time Point

| | | | Serum EV68-228-N Concentrations | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose<br>Coho<br>rt | Particip<br>ant ID | Pre-<br>Infusion<br>(-15 min) | End of<br>Infusion<br>(+ 5 min) | 1-hour<br>(± 15 min) | 3-hour<br>(± 15 min) | 5-hour<br>(± 15 min) | 24-hour<br>(± 3 hr) | 48-hour<br>(± 3 hr) | 7-day<br>(± 1 day) | 14-day<br>(± 2 day) | 28-day<br>(± 3 day) | 60-day<br>(± 7 day) | 90-day<br>(± 14 day) | 120-day<br>(± 14 day) |
| 3<br>mg/k | XXXXX<br>XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXX<br>XX.XXX |
| g<br>EV68<br>-228-<br>N | | | | | | | | | | | | | | |
| 10mg<br>/kg | XXXXX<br>XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXX<br>XX.XXX |
| EV68<br>-228-<br>N | | | | | | | | | | | | | | |
| 30<br>mg/k | XXXXX<br>XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX |
| g<br>EV68<br>-228-<br>N | | are reported i | | | | | | | | | | | | |

Note: Concentrations are reported in units of ng/mL.

**Table 78:** Summary Statistics of Serum EV68-228-N Concentrations by Time Point

| | Sum | | | | | | Serum EV | 68-228-N Con | centrations | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose<br>Coh<br>ort | mary<br>Statis<br>tics | Pre-<br>Infusion<br>(-15 min) | End of<br>Infusion<br>(+ 5 min) | 1-hour<br>(± 15 min) | 3-hour<br>(± 15 min) | 5-hour<br>(± 15 min) | 24-hour<br>(± 3 hr) | 48-hour<br>(± 3 hr) | 7-day<br>(± 1 day) | 14-day<br>(± 2 day) | 28-day<br>(± 3 day) | 60-day<br>(± 7 day) | 90-day<br>(± 14 day) | 120-day<br>(± 14 day) |
| 3 | N | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| mg/k<br>g<br>EV6<br>8-<br>228- | Mean<br>(SD) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) |
| N | Min,<br>Max | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX |
| | Geom<br>etric<br>Mean | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX |
| | CV% | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 10m | N | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| g/kg<br>EV6<br>8-<br>228-<br>N | Mean<br>(SD) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) |
| | Min,<br>Max | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX |
| | Geom<br>etric<br>Mean | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX |
| | CV% | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| 30 | N | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| mg/k<br>g<br>EV6<br>8- | Mean<br>(SD) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) | XXXXXX<br>.XXX<br>(XXXXX<br>X.XXX) |

Table 78: Summary Statistics of Serum EV68-228-N Concentrations by Time Point (continued)

| | Sum | | | | | | Serum EV | 68-228-N Con | centrations | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose<br>Coh<br>ort | mary<br>Statis<br>tics | Pre-<br>Infusion<br>(-15 min) | End of<br>Infusion<br>(+ 5 min) | 1-hour<br>(± 15 min) | 3-hour<br>(± 15 min) | 5-hour<br>(± 15 min) | 24-hour<br>(± 3 hr) | 48-hour<br>(± 3 hr) | 7-day<br>(± 1 day) | 14-day<br>(± 2 day) | 28-day<br>(± 3 day) | 60-day<br>(± 7 day) | 90-day<br>(± 14 day) | 120-day<br>(± 14 day) |
| 228-<br>N | Min,<br>Max | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX | XXXXXX<br>.XXX,<br>XXXXXX<br>.XXX |
| | Geom<br>etric<br>Mean | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX | XXXXXX<br>.XXX |
| | CV% | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Notes: N=Number of participants in the PK Population. Concentrations are reported in units of ng/mL.

## Table 79: Individual Statistics of Noncompartmental Serum PK Parameters by Dose Cohort

| Dose Cohort | Participant ID | AUC₀-∞<br>(ng*h/mL) | AUC <sub>0-last</sub><br>(ng*h/mL) | AUC <sub>0-48</sub><br>(ng*h/mL) | C <sub>max</sub> (ng/mL) | T <sub>max</sub> (h) | t <sub>1/2</sub> (h) | CL<br>(L/h) | V <sub>z</sub> (h) |
|---|---|---|---|---|---|---|---|---|---|
| 3 mg/kg EV68-228-N | XXXXXXXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |
| 10 mg/kg EV68-228-N | XXXXXXXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |
| 30 mg/kg EV68-228-N | XXXXXXXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |

Table 80: Summary Statistics of Noncompartmental Serum PK Parameters by Dose Cohort

| Dose<br>Cohort | Summary<br>Statistics | AUC₀-∞<br>(ng*h/mL) | AUC <sub>0-last</sub><br>(ng*h/mL) | AUC <sub>0-48</sub><br>(ng*h/mL) | C <sub>max</sub><br>(ng/mL) | T <sub>max</sub> (h) | t <sub>1/2</sub> (h) | CL<br>(L/h) | V <sub>z</sub> (L) |
|---|---|---|---|---|---|---|---|---|---|
| 3 mg/kg | N | XX | XX | XX | XX | XX | XX | XX | XX |
| EV68-<br>228-N | Mean (SD) | XXXXXX.XXX<br>(XXXXXXXXXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXX.X<br>(XXX.X) | XXX.X<br>(XXX.X) | XXX.X<br>(XXX.X) | XXXX.X<br>(XXXX.X) |
| | Min, Max | XXXXXX.XXX,<br>XXXXXX.XXX | XXXXXX.XXX,<br>XXXXXXXXX | XXXXXX.XXX,<br>XXXXXXXXX | XXXXXX.XXX,<br>XXXXXXXXX | XXX.X,<br>XXX.X | XXX.X,<br>XXX.X | XXX.X,<br>XXX.X | XXXX.X,<br>XXXX.X |
| | Geometric<br>Mean | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |
| | CV% | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |
| 10 mg/kg | N | XX | XX | XX | XX | XX | XX | XX | XX |
| EV68-<br>228-N | Mean (SD) | XXXXXX.XXX<br>(XXXXXXXXXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXX.X<br>(XXX.X) | XXX.X<br>(XXX.X) | XXX.X<br>(XXX.X) | XXXX.X<br>(XXXX.X) |
| | Min, Max | XXXXXX.XXX,<br>XXXXXXXXX | XXXXXX.XXX,<br>XXXXXXXXX | XXXXXX.XXX,<br>XXXXXXXXX | XXXXXX.XXX,<br>XXXXXXXXX | XXX.X,<br>XXX.X | XXX.X,<br>XXX.X | XXX.X,<br>XXX.X | XXXX.X,<br>XXXX.X |
| | Geometric<br>Mean | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |
| | CV% | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |
| 30 mg/kg | N | XX | XX | XX | XX | XX | XX | XX | XX |
| EV68-<br>228-N | Mean (SD) | XXXXXX.XXX<br>(XXXXXXXXXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXXXXX.XXX<br>(XXXXXX.XXX) | XXX.X<br>(XXX.X) | XXX.X<br>(XXX.X) | XXX.X<br>(XXX.X) | XXXX.X<br>(XXXX.X) |
| | Min, Max | XXXXXX.XXX,<br>XXXXXXXXX | XXXXXX.XXX,<br>XXXXXXXXX | XXXXXX.XXX,<br>XXXXXX.XXX | XXXXXX.XXX,<br>XXXXXXXXX | XXX.X,<br>XXX.X | XXX.X,<br>XXX.X | XXX.X,<br>XXX.X | XXXX.X,<br>XXXX.X |
| | Geometric<br>Mean | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |
| | CV% | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXXXXX.XXX | XXX.X | XXX.X | XXX.X | XXXX.X |

Note: N=Number of participants in the PK Population used to calculate the summary statistics.

# APPENDIX 2. FIGURE MOCK-UPS

| Figure 1: | CONSORT Flow Diagram | 116 |
|---|---|---|
| Figure 2: | Reverse Cumulative Distribution of ADAs by Time Point and Dose Cohort | 117 |
| Figure 3: | Maximum Severity of Solicited Symptoms per Participant by Day Post Treatment | 118 |
| Figure 4: | Frequency of Related Adverse Events by MedDRA System Organ Class and Severity | 119 |
| Figure 5: | Incidence of Related Adverse Events by MedDRA System Organ Class and Maximum Severity | 120 |
| Figure 6: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort –Creatinine | 121 |
| Figure 7: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort – Total Bilirubin | 121 |
| Figure 8: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort – ALT | 121 |
| Figure 9: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort – Hemoglobin | 121 |
| Figure 10: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort – WBC | 121 |
| Figure 11: | Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort – Platelets | 121 |
| Figure 12: | Linear Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 3 mg/kg EV68-228-N Dose Cohort | 122 |
| Figure 13: | Linear Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 10 mg/kg EV68-228-N Dose Cohort | 122 |
| Figure 14: | Linear Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 30 mg/kg EV68-228-N Dose Cohort | |
| Figure 15: | Semilogarithmic Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 3 mg/kg EV68-228-N Dose Cohort | 123 |
| Figure 16: | Semilogarithmic Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 10 mg/kg EV68-228-N Dose Cohort | |
| Figure 17: | Semilogarithmic Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 30 mg/kg EV68-228-N Dose Cohort | 123 |
| Figure 18: | Linear Plot of Mean ± SD of EV68-228-N Serum Concentration by Nominal Time and Dose Cohort | |
| Figure 19: | Semilogarithmic Plot of Mean ± SD of EV68-228-N Serum Concentration by Nominal Time and Dose Cohort | 125 |

#### 10.1 Disposition of Participants

Figure 1: CONSORT Flow Diagram



# 14.2.2 Immunogenicity Response Figures by Measure, Treatment/Vaccination, and Time Point

Figure 2: Reverse Cumulative Distribution of ADAs by Time Point and Dose Cohort



#### 14.3.1.1 Solicited Adverse Events

Figure 3: Maximum Severity of Solicited Symptoms per Participant by Day Post Treatment [Implementation Note: Separated panels for each Dose Cohort.]



#### 14.3.1.2 Unsolicited Adverse Events

Figure 4: Frequency of Related Adverse Events by MedDRA System Organ Class and Severity



Figure 5: Incidence of Related Adverse Events by MedDRA System Organ Class and Maximum Severity



#### 14.3.5 Displays of Laboratory Results

Figure 6: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort - Creatinine

[Implementation Note: This plot is just an illustration. Each dose cohort will have a separated panel, plot will not be separated by gender.]



Figures with similar format:

- Figure 7: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort Total Bilirubin
- Figure 8: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort ALT
- Figure 9: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort Hemoglobin
- Figure 10: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort WBC
- Figure 11: Laboratory Results by Scheduled Visits: Mean Changes from Baseline by Laboratory Parameter, and Dose Cohort Platelets

Figure 12: Linear Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 3 mg/kg EV68-228-N Dose Cohort

[Implementation Note: Update "Participant" and numbers in the legend to the "Participant ID" and use USUBJID (or equivalent). Update the LLOQ to the appropriate value based on the assay. The vertical axis label should be "EV68-228-N Concentration (Units)" where units are updated accordingly, and the horizontal axis label should be updated to days based on the protocol specified sampling scheme. Samples that are <LLOQ should not be plotted.]



Figures with same format:

Figure 13: Linear Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 10 mg/kg EV68-228-N Dose Cohort

Figure 14: Linear Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 30 mg/kg EV68-228-N Dose Cohort

Figure 15: Semilogarithmic Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 3 mg/kg EV68-228-N Dose Cohort

[Implementation Note: Update "Participant" and numbers in the legend to the "Participant ID" and use USUBJID (or equivalent). Update the LLOQ to the appropriate value based on the assay. The vertical axis label should be "EV68-228-N Concentration (Units)" where units are updated accordingly, and the horizontal axis label should be updated to days based on the protocol specified sampling scheme. Samples that are <LLOQ should not be plotted]



Figures with similar format:

Figure 16: Semilogarithmic Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 10 mg/kg EV68-228-N Dose Cohort

Figure 17: Semilogarithmic Plot of EV68-228-N Serum Concentration Profiles by Nominal Time – 30 mg/kg EV68-228-N Dose Cohort

Figure 18: Linear Plot of Mean  $\pm$  SD of EV68-228-N Serum Concentration by Nominal Time and Dose Cohort

[Implementation Note: Update "Units" accordingly as well as the actual LLOQ value. Samples that are <LLOQ should not be plotted]



Figure 19: Semilogarithmic Plot of Mean  $\pm$  SD of EV68-228-N Serum Concentration by Nominal Time and Dose Cohort

[Implementation Note: Update "Units" accordingly as well as the actual LLOQ value. Samples that are <LLOQ should not be plotted.]



# APPENDIX 3. LISTINGS MOCK-UPS

| Listing 1: | 16.1.6: Listing of Participants Receiving Investigational Product | 127 |
|---|---|---|
| Listing 2: | 16.2.1: Early Terminations or Discontinued Participants | 128 |
| Listing 3: | 16.2.2.1: Participant-Specific Protocol Deviations | 129 |
| Listing 4: | 16.2.2.2: Non-Participant-Specific Protocol Deviations | 130 |
| Listing 5: | 16.2.3: Participants Excluded from Analysis Populations | 131 |
| Listing 6: | 16.2.4.1: Demographic Data | 132 |
| Listing 7: | 16.2.4.2: Pre-Existing and Concurrent Medical Conditions | 133 |
| Listing 8: | 16.2.5: Compliance Data | 134 |
| Listing 9: | 16.2.5: Infusion Interruptions | 135 |
| Listing 10: | 16.2.6: Immunogenicity Response Data | 136 |
| Listing 11: | 16.2.7.1: Solicited Adverse Events | 137 |
| Listing 12: | 16.2.7.3: Unsolicited Adverse Events | 138 |
| Listing 13: | 16.2.8.1: Clinical Laboratory Results – Chemistry | 139 |
| Listing 14: | 16.2.8.2: Clinical Laboratory Results – Hematology | 140 |
| Listing 15: | 16.2.9.1: Vital Signs | 141 |
| Listing 16: | 16.2.9.2: Abnormal Physical Exam Findings | 142 |
| Listing 17: | 16.2.10: Concomitant Medications | 143 |
| Listing 18: | 16.2.11.1: Pregnancy Reports – Maternal Information | 144 |
| Listing 19: | 16.2.11.2: Pregnancy Reports – Gravida and Para | 145 |
| Listing 20: | 16.2.11.3: Pregnancy Reports – Live Birth Outcomes | 146 |
| Listing 21: | 16.2.11.4: Pregnancy Reports – Still Birth Outcomes | 147 |
| Listing 22: | 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes | 148 |
| Listing 23: | 16.2.9.4: Listing of Individual ECG Parameters | 149 |
| Listing 24: | 16.2.9.4: Listing of ECG Overall Interpretation and Comments | 150 |
| Listing 25. | 16.2.9.4: Participant Level Drug Concentrations | 151 |

## **Listing 1:** 16.1.6: Listing of Participants Receiving Investigational Product

(not included in SAP, but this is a placeholder for the CSR)

## 16.2 Database Listings by Participant

## **16.2.1 Discontinued Participants**

## **Listing 2:** 16.2.1: Early Terminations or Discontinued Participants

[Implementation Note: Data need to be sorted by Dose Cohort, Participant ID, Category.]

| Dose Cohort | Participant ID | Category | Reason for Early Termination or Treatment Discontinuation | Study Day |
|---|---|---|---|---|

#### **16.2.2 Protocol Deviations**

#### **Listing 3:** 16.2.2.1: Participant-Specific Protocol Deviations

[Implementation Notes:

- 1. Treatment group is the randomized treatment group.
- 2. Sort order will be by Treatment Group, Subject ID, Deviation Number.
- 3. Deviation description column will contain all subfields (comments) concatenated together.]

| Dose<br>Cohort | Participant<br>ID | DV<br>Number | Study Day | Deviation<br>Classification | Deviation<br>Description | Deviation<br>Category | Reason for<br>Deviation | Deviation<br>Resulted in<br>AE? | Deviation Resulted in<br>Participant<br>Termination? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | Major/Minor | | | | | | | |

#### **Listing 4:** 16.2.2.2: Non-Participant-Specific Protocol Deviations

[Implementation Notes:

- 1. Sort order will be by Site Name, Start Date
- 2. In the Deviation column concatenate any specified fields
- 3. In the Reason for Deviation column concatenate any specified fields.]

| Site | Start<br>Date | Deviation | End Date | Reason for<br>Deviation | Deviation Resulted<br>in Participant<br>Termination? | Deviation<br>Affected<br>Product<br>Stability? | Deviation<br>Category | Deviation<br>Classification? | Deviation<br>Resolution | Comments |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Major/Minor | | |

#### 16.2.3 Participants Excluded from the Efficacy Analysis

## **Listing 5:** 16.2.3: Participants Excluded from Analysis Populations

| Dose Cohort | Participant ID | Analyses in which<br>Participant is Included | Analyses from which<br>Participant is Excluded | Results Available? | Reason Participant Excluded |
|---|---|---|---|---|---|
| | | [e.g., Safety, mITT, PK, Imm] | [e.g., Safety, mITT, PK, Imm, Day x] | | |

Note: "Yes" in the "Results available" column indicates that available data were removed from the analysis. "No" indicates that no data were available for inclusion in the analysis.

## 16.2.4 Demographic Data

# Listing 6: 16.2.4.1: Demographic Data

| Dose Cohort | Participant ID | Sex | Sex Assigned at Birth | Gender Identity | Age at Enrollment (years) | Ethnicity | Race |
|---|---|---|---|---|---|---|---|

# Listing 7: 16.2.4.2: Pre-Existing and Concurrent Medical Conditions

| <b>Dose Cohort</b> | t Participant ID MH Number Medic | Medical History Term | <b>Condition Start Day</b> | <b>Condition End Day</b> | MedDRA System Organ Class | MedDRA Preferred Term |
|---|---|---|---|---|---|---|

#### 16.2.5 Compliance and/or Drug Concentration Data (if available)

## Listing 8: 16.2.5: Compliance Data

[Implementation Note: For planned doses that did not occur, the date and time columns for those doses will be "not dosed." Sort Order: Dose Cohort, Participant ID.]

| Dose Cohort | Participant ID | Dose Date | Infusion<br>Administration Site | Infusion Start<br>Time | Volume to be Infused (mL) | Total Volume<br>Administered<br>(mL) | Planned Volume<br>Administered? | Infusion End Time |
|---|---|---|---|---|---|---|---|---|
| | | ddMMMyyyy | Left Arm/<br>Right Arm | hh:mm | | | Yes/No | hh:mm |

#### **Listing 9:** 16.2.5: Infusion Interruptions

[Implementation Note: For planned doses that did not occur, the date and time columns for those doses will be "not dosed." Sort Order: Dose Cohort, Participant ID.]

| Dose<br>Cohort | Participant<br>ID | Interruption<br>Number | Interruption<br>Time<br>(hh:mm) | Reason<br>Infusion<br>Interrupted | Volume of IP Infused<br>Prior to Interruption<br>(mL) | Infusion<br>Restarted? | Restart<br>Time<br>(hh:mm) | Interrupted<br>Again? | Infusion<br>Discontinued? | Reason for<br>Discontinuation | Infusion<br>Completed? |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | Yes/No | | Yes/No | Yes/No | | Yes/No |

#### 16.2.6 Individual Efficacy/Immunogenicity Response Data

## Listing 10: 16.2.6: Immunogenicity Response Data

[Implementation note:

For Screening Result, it could be NEG/PPS/NRR, which means Negative/Potential Positive/No Recorded Result.

For Confirmatory Result, it will report the results for samples that were potential positive in screening. Null for screening negative, NRR for screening NRR.

For Titer, reports titer results for samples that confirmed positive in confirmatory results. NULL for negative confirmatory results. NRR for NRR confirmatory results.]

| Dose<br>Cohort | Participant ID | Planned Time<br>Point | Actual Study Day | Screening Results <sup>a</sup> | Confirmatory Results <sup>b</sup> | Titer <sup>c</sup> | Comment |
|---|---|---|---|---|---|---|---|
| | | | | NEG | NULL | NA | |
| | | | | PPS | NEG | NULL | |
| | | | | PPS | POS | xxxxx | |
| | | | | PPS | NRR | NRR | |
| | | | | NRR | NRR | NA | |

<sup>&</sup>lt;sup>a</sup>The ADA screening assay result could be Negative (NEG), Potential Positive (PPS), or No Recorded Result (NRR).

<sup>&</sup>lt;sup>b</sup>The ADA confirmatory assay was performed for those specimens with a PPS screening result. The confirmatory result could be Negative (NEG), Positive (POS), or No Result Recorded (NNR). If screening result is NEG, then the confirmatory result is NRR.

<sup>&</sup>lt;sup>c</sup>The ADA titer assay was reported for those specimens with a POS confirmatory result. If confirmatory result is NEG, then the titer is NULL. If confirmatory result is NRR, then the titer is NRR. If the screen result was NEG or NRR, then the titer is NA.

#### 16.2.7 Adverse Events

**Listing 11: 16.2.7.1: Solicited Adverse Events** 

| Dose Cohort | Participant ID | Post Dose Day | Assessment <sup>a</sup> | Symptom | Severity | Attributed to Alternate Etiology? | Alternate Etiology |
|---|---|---|---|---|---|---|---|
| | | | MA | | | | |
| | | | Clinic | | | | |

<sup>&</sup>lt;sup>a</sup> MA = Data reported by participant on the Memory Aid and reviewed by clinic staff and reported in Solicited Events eCRF.

Note: Clinic = Data collected by clinic staff during physical exam or symptom assessment (treatment administration record, in-clinic assessment, etc.).

#### **Listing 12:** 16.2.7.3: Unsolicited Adverse Events

| Adverse Event | No. of<br>Days Post<br>Dose<br>(Duration) | Severity | SAE? | MAAE/<br>NOCMC/<br>UP? | Relationship<br>to Study<br>Treatment | In Not<br>Related,<br>Alternative<br>Etiology | Action<br>Taken<br>with<br>Study<br>Treatment | Participant<br>Discontinued<br>Due to AE | Outcome | MedDRA<br>System Organ Class | MedDRA<br>High Level<br>Group<br>Term | MedDRA<br>Preferred<br>Term |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Dose Cohort, Par | rticipant ID, A | AE Number | : | | | | | | | | | |
| Comments: | | | | | | | | | | | | |
| Dose Cohort, Par | Dose Cohort, Participant ID, AE Number: | | | | | | | | | | | |
| Comments: | | | | | • | | | | • | | , | |

Note: For additional details about SAEs, see section 14.3.2.

## 16.2.8 Individual Laboratory Measurements

# **Listing 13:** 16.2.8.1: Clinical Laboratory Results – Chemistry

| Dose Cohort | Participant ID | Planned Time<br>Point | Actual<br>Study Day | Laboratory Parameter (Units) | Result (Severity<br>Grade) | Reference Range<br>Low | Reference Range<br>High | Comments |
|---|---|---|---|---|---|---|---|---|

# **Listing 14:** 16.2.8.2: Clinical Laboratory Results – Hematology

| Dose Cohort | Participant ID | Planned Time<br>Point | Actual Study<br>Day | Laboratory Parameter (Units) | Result<br>(Severity Grade) | Reference Range<br>Low | Reference Range<br>High | Comments |
|---|---|---|---|---|---|---|---|---|

#### 16.2.9 Vital Signs and Physical Exam Findings

#### Listing 15: 16.2.9.1: Vital Signs

[Implementation note: The BMI is calculated with height at screening and weight at day prior to dosing. – do NOT report the Screening BMI. Will be consistent with the summarized table (Table 11 and 13)]

| Dose<br>Cohort | Participant<br>ID | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Time of<br>Assessment<br>(hh:mm) | Replicate | Temperature (°C) | Systolic<br>Blood<br>Pressure<br>(mmHg) | Diastolic<br>Blood<br>Pressure<br>(mmHg) | Pulse<br>(beats/min) | SpO2<br>(%) | Height (cm) | Weight<br>(kg) | BMI<br>(kg/m2) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

## Listing 16: 16.2.9.2: Abnormal Physical Exam Findings

| Dose Cohort | Participant ID | Planned Time Point | Actual Study Day | Body System | Abnormal Finding | Reported as an AE? |
|---|---|---|---|---|---|---|
| | | | | | | No /Yes, solicited AE. Specify solicited AE: /Yes, unsolicited AE, AE description, AE # |

#### **16.2.10** Concomitant Medications

# **Listing 17: 16.2.10: Concomitant Medications**

| Dose<br>Cohort | Participant<br>ID | CM<br>Number | Medication | Medication Start Day | Medication End Day | Indication | Taken for an AE? | Taken for a condition on<br>Medical History?<br>(MH Description; MH Number) | ATC Level 1<br>(ATC Level 2) |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | No /Yes, solicited AE. Specify solicited AE: /Yes, unsolicited AE, AE description, AE # | | |

#### 16.2.11 Pregnancy Reports

## **Listing 18:** 16.2.11.1: Pregnancy Reports – Maternal Information

| Dose<br>Cohort | Participant<br>ID | Pregnancy<br>Number | Study Day Corresponding to Estimated Date of Conception | Source of<br>Maternal<br>Information | Pregnancy<br>Status | Mother's<br>Pre-<br>Pregnancy<br>BMI | Mother's<br>Weight<br>Gain<br>During<br>Pregnancy | Tobacco, Alcohol, or Drug Use During Pregnancy? | Medications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During<br>Pregnancy? | Maternal<br>Complications<br>During Labor,<br>Delivery, or Post-<br>Partum? |
|---|---|---|---|---|---|---|---|---|---|---|---|

Notes: Maternal Complications are included in the Adverse Event listing. Medications taken during pregnancy are included in the Concomitant Medications Listing.

Listing 19: 16.2.11.2: Pregnancy Reports – Gravida and Para

| | | | | Live Births | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Participant<br>ID | Pregnancy<br>Number | Gravida | Extremely<br>PB <sup>a</sup> | Very<br>Early<br>PB <sup>a</sup> | Early<br>PB <sup>a</sup> | Late<br>PB <sup>a</sup> | Early<br>TB <sup>a</sup> | Full<br>TB <sup>b</sup> | Late<br>TB <sup>b</sup> | Post<br>TB <sup>b</sup> | Still<br>Births | Spontaneous<br>Abortion/<br>Miscarriage | Elective<br>Abortions | Therapeutic<br>Abortions | Major<br>Congenital<br>Anomaly<br>with<br>Previous<br>Pregnancy? |

Note: Gravida includes the current pregnancy, para events do not.

a Preterm Birth
b Term Birth

## **Listing 20:** 16.2.11.3: Pregnancy Reports – Live Birth Outcomes

| Participant<br>ID | Pregnancy<br>Number | Fetus<br>Number | Pregnancy<br>Outcome (for<br>this Fetus) | Fetal Distress<br>During Labor<br>and Delivery? | Delivery<br>Method | Gestational<br>Age at Live<br>Birth | Size for<br>Gestational<br>Age | Apgar<br>Score, 1<br>minute | Apgar<br>Score, 5<br>minutes | Cord<br>pH | Congenital<br>Anomalies? | Illnesses/<br>Hospitalizations<br>within 1 Month of<br>Birth? |
|---|---|---|---|---|---|---|---|---|---|---|---|---|

Note: Congenital Anomalies are included in the Adverse Event listing.

## **Listing 21:** 16.2.11.4: Pregnancy Reports – Still Birth Outcomes

| Participant<br>ID | Date of<br>Initial<br>Report | Fetus<br>Number | Pregnancy<br>Outcome (for<br>this Fetus) | Fetal Distress<br>During Labor<br>and Delivery? | Delivery<br>Method | Gestational<br>Age at Still<br>Birth | Size for<br>Gestational<br>Age | Cord pH | Congenital Anomalies? | Autopsy<br>Performed? | If Autopsy,<br>Etiology for Still<br>Birth Identified? |
|---|---|---|---|---|---|---|---|---|---|---|---|

## **Listing 22:** 16.2.11.5: Pregnancy Reports – Spontaneous, Elective, or Therapeutic Abortion Outcomes

| Participant<br>ID | Date of Initial<br>Report | Fetus Number | Pregnancy Outcome<br>(for this Fetus) | Gestational Age at<br>Termination | Abnormality in Product of Conception? | Reason for Therapeutic<br>Abortion |
|---|---|---|---|---|---|---|

#### 16.2.9 Individual ECG Results

# **Listing 23:** 16.2.9.4: Listing of Individual ECG Parameters

[Implementation Note: This listing includes all ECG assessments, scheduled and unscheduled. Sort order: Dose Cohort, Participant ID, Parameter, Date of Assessment, Time of Assessment.]

| Dose<br>Cohort | Participant<br>ID | Planned<br>Time Point | Actual<br>Study<br>Day | Assessment | | Right Bundle<br>Branch Block | | Advanced<br>A-V Heart<br>Block | Non-<br>sinus<br>Rhythm | Pathologic<br>Q wave<br>Abnormalities | Significant<br>ST-T Wave<br>Changes | Prolonged<br>QTc<br>Interval | Other |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Baseline | | | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | |
| | | 1 hour after infusion | | | | | | | | | | | |
| | | Day 2 | | | | | | | | | | | |

#### Listing 24: 16.2.9.4: Listing of ECG Overall Interpretation and Comments

[Implementation Note: This listing includes all ECG assessments, scheduled and unscheduled. Sort order: Dose Cohort, Participant ID, Parameter, Date of Assessment, Time of Assessment.

When Overall interpretation is normal, or abnormal NCS, then it will be 'NA' for column 'clinically significant']

| Dose<br>Cohort | Participant<br>ID | Planned<br>Time<br>Point | Actual<br>Study<br>Day | Time of<br>Assessment<br>(hh:mm) | Any Immediate Issues | Overall Interpretation | Clinically Significant? | Comments |
|---|---|---|---|---|---|---|---|---|
| | | Baseline | | | No/Yes, specify | Normal | NA | |
| | | 1 hour<br>after<br>infusion | | | No/Yes, specify | Normal/Abnormal NCS<br>/Abnormal CS | No/Yes, specify | |
| | | Day 2 | | | No/Yes, specify | Normal/Abnormal<br>NCS/Abnormal CS | No/Yes, specify | |

**Listing 25:** 16.2.9.4: Participant Level Drug Concentrations

| Participant ID | Nominal<br>Time Point<br>(hours) | Actual Time pPoint (hours) | Sample Collected<br>Within Time Window | EV68-228-N<br>Concentration<br>(ng/mL) | Used in λz<br>Calculation? | Excluded from PK Analysis | Reason For Exclusion from PK Analysis |
|---|---|---|---|---|---|---|---|
| XXXXXXXX | Pre-Infusion | Pre-Infusion | Yes | 0.00 | No | No | N/A |
| XXXXXXXX | 0 | 0.067 | Yes | XXXX.XX | No | No | N/A |
| XXXXXXXX | 1 | 1.2 | Yes | XXXX.XX | No | No | N/A |
| XXXXXXXX | 3 | 2.9 | Yes | XXXX.XX | No | No | N/A |
| XXXXXXXX | 5 | 5.5 | No | XXXX.XX | No | No | N/A |
| XXXXXXXX | 24 | - | - | XXXX.XX | No | No | N/A |
| XXXXXXXX | 48 | 51.25 | No | XXXX.XX | No | No | N/A |
| XXXXXXXX | 168 | 180.06 | Yes | XXXX.XX | No | No | N/A |
| XXXXXXXX | 336 | 330.25 | Yes | XXXX.XX | No | No | N/A |
| XXXXXXXX | 672 | 700.5 | Yes | XXXX.XX | Yes | No | N/A |
| XXXXXXXX | 1440 | 1442.1 | Yes | XXXX.XX | Yes | No | N/A |
| XXXXXXXX | 2160 | 2159.33 | Yes | BQL* | Yes | No | N/A |
| XXXXXXXX | 2880 | 2866 | Yes | BQL | No | Yes | BQL treated as missing |
| XXXXXXXX | Pre-Infusion | Pre-Infusion | Yes | 0 | No | No | N/A |
| XXXXXXXX | Pre-Infusion | Pre-Infusion | Yes | 0 | No | No | N/A |
| | XXXXXXXX XXXXXXXX XXXXXXXX XXXXXXXX XXXX | Participant ID Time Point (hours) XXXXXXXXX Pre-Infusion XXXXXXXXX 0 XXXXXXXXX 1 XXXXXXXXX 3 XXXXXXXXX 5 XXXXXXXXX 24 XXXXXXXXX 168 XXXXXXXXX 336 XXXXXXXXX 672 XXXXXXXXX 2160 XXXXXXXXX 2880 XXXXXXXXX Pre-Infusion | Participant ID Time Point (hours) pPoint (hours) XXXXXXXXX Pre-Infusion Pre-Infusion XXXXXXXXX 0 0.067 XXXXXXXXX 1 1.2 XXXXXXXXX 3 2.9 XXXXXXXXX 5 5.5 XXXXXXXXX 24 - XXXXXXXXX 168 180.06 XXXXXXXXX 336 330.25 XXXXXXXXX 672 700.5 XXXXXXXXX 1440 1442.1 XXXXXXXXX 2160 2159.33 XXXXXXXXX 2880 2866 XXXXXXXXX Pre-Infusion Pre-Infusion | Participant ID Time Point (hours) pPoint (hours) Sample Collected Within Time Window XXXXXXXXX Pre-Infusion Yes XXXXXXXXX 0 0.067 Yes XXXXXXXXX 1 1.2 Yes XXXXXXXXX 3 2.9 Yes XXXXXXXXX 5 5.5 No XXXXXXXXX 24 - - XXXXXXXXX 48 51.25 No XXXXXXXXX 168 180.06 Yes XXXXXXXXX 336 330.25 Yes XXXXXXXXX 672 700.5 Yes XXXXXXXXX 2160 2159.33 Yes XXXXXXXXX 2880 2866 Yes XXXXXXXXX Pre-Infusion Pre-Infusion Yes | Participant ID Time Point (hours) pPoint (hours) Sample Collected Within Time Window Concentration (ng/mL) XXXXXXXXX Pre-Infusion Pres 0.00 XXXXXXXXX 0 0.067 Yes XXXXXXX XXXXXXXXX 1 1.2 Yes XXXXXXXX XXXXXXXXX 3 2.9 Yes XXXXXXXX XXXXXXXXX 5 5.5 No XXXXXXXX XXXXXXXXX 24 - - XXXXXXXX XXXXXXXXX 48 51.25 No XXXXXXXX XXXXXXXXX 168 180.06 Yes XXXXXXXX XXXXXXXXX 336 330.25 Yes XXXXXXXX XXXXXXXXX 672 700.5 Yes XXXXXXXX XXXXXXXXX 2160 2159.33 Yes BQL* XXXXXXXXX Pre-Infusion Pre-Infusion Yes 0 | Participant ID Time Point (hours) pPoint (hours) Sample Collected Within Time Window Concentration (ng/mL) Used in λz Calculation? XXXXXXXXX Pre-Infusion Yes 0.00 No XXXXXXXXX 0 0.067 Yes XXXXXXXX No XXXXXXXXX 1 1.2 Yes XXXXXXXX No XXXXXXXXX 3 2.9 Yes XXXXXXXX No XXXXXXXXX 5 5.5 No XXXXXXXX No XXXXXXXXX 24 - - XXXXXXXX No XXXXXXXXX 48 51.25 No XXXXXXXX No XXXXXXXXX 168 180.06 Yes XXXXXXXX No XXXXXXXXX 336 330.25 Yes XXXXXXXX No XXXXXXXXX 672 700.5 Yes XXXXXXXX Yes XXXXXXXXX 1440 1442.1 Yes BQL No XXXXXXXXX 2880 2866 Yes | Participant ID Time Point (hours) pPoint (hours) Sample Collected Within Time Window Concentration (ng/mL) Used in \( \frac{\pi}{2} \) Excluded from PK Analysis XXXXXXXXX Pre-Infusion Yes 0.00 No No XXXXXXXXX 0 0.067 Yes XXXXXXX No No XXXXXXXXX 1 1.2 Yes XXXXXXX No No XXXXXXXXX 3 2.9 Yes XXXXXXXX No No XXXXXXXXX 5 5.5 No XXXXXXXX No No XXXXXXXXX 24 - - XXXXXXXX No No XXXXXXXXX 48 51.25 No XXXXXXXX No No XXXXXXXXX 168 180.06 Yes XXXXXXXX No No XXXXXXXXX 336 330.25 Yes XXXXXXXX No No XXXXXXXXX 672 700.5 Yes XXXXXXXX Yes No |

<sup>\*</sup> Denotes a sample that was reported as BQL but was imputed as LLOQ/2 because it was necessary to compute  $\lambda z$  during the noncompartmental analysis. Note: Missing actual time points were imputed as the nominal time point for the purpose of analysis.